CLINICAL TRIAL: NCT03000569
Title: A Phase 2, Two-Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of SAGE-217 in Subjects With Parkinson's Disease
Brief Title: A Study to Evaluate SAGE-217 in Participants With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 217-PRK-201
Record Dates: First submitted 2016-11-28; First posted 2016-12-22 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's
MeSH Terms: conditions — Parkinson Disease | interventions — zuranolone; Levodopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: Antiparkinsonian Agent(s) Followed by SAGE-217 (Experimental): Participants on a stable morning dose of levodopa (including carbidopa-levodopa) as antiparkinsonian agent(s) from Days 1 to 3, stopped levodopa and received SAGE-217 at a dose of 30 mg per day, oral solution, for Days 4 to 7 in the morning with food. Stable doses of other antiparkinsonian agents and dose reductions in SAGE-217 were allowed between Days 1 to 7. Participants resumed stable morning dose of levodopa from Days 8 to 14.
  Interventions: Drug: SAGE-217; Drug: Levodopa
- Part B: Antiparkinsonian Agent(s) + SAGE-217 (Experimental): Participants on a stable dose of antiparkinsonian agent(s) received SAGE-217, up to 30 mg per day, capsules, for Days 1 to 7 in the evening with food.
  Interventions: Drug: SAGE-217; Drug: Antiparkinsonian Agent(s)

INTERVENTIONS:
Drug: SAGE-217
Drug: Levodopa — Levodopa (including carbidopa-levodopa) administered as antiparkinsonian agent(s).
  Arms: Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Drug: Antiparkinsonian Agent(s) — Antiparkinsonian agent(s) were administered as a clinical practice as standard of care, which includes levodopa (i.e. levodopa/carbidopa) or dopamine agonists or catechol-O-methyltransferase (COMT) inhibitors or monoamine oxidase (BMAO-B) inhibitors.
  Arms: Part B: Antiparkinsonian Agent(s) + SAGE-217

SUMMARY:
This study assesses the safety, tolerability, pharmacokinetics and efficacy of SAGE-217 in 29 participants with moderate to severe Parkinson's Disease.

DETAILED DESCRIPTION:
Part A of the study is an open-label design with dosing of Levodopa for 3 days followed by SAGE-217 for 4 days.

Part B of the study is an open-label design with evening dosing of SAGE-217 for 7 days as an adjunct to antiparkinsonian agent(s).

This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of idiopathic Parkinson's Disease (Hoehn and Yahr Stage 2 or Stage 3) with a duration of less than 7 years prior to screening [Part A]
* Participant has a diagnosis of idiopathic Parkinson's Disease (Hoehn and Yahr Stage 1-4, assessed during the "on" period) [Part B]
* Participant is on a stable dose (at least 1 month prior to baseline visit) of an antiparkinsonian agent and is willing to remain on this dose for the duration of the study

Exclusion Criteria:

* Participant has early (Hoehn and Yahr Stage 1) or advanced (Hoehn and Yahr Stage 4 or Stage 5) Parkinson's Disease [Part A]
* Participant has advanced (Hoehn and Yahr Stage 5) Parkinson's Disease [Part B]
* Participant with presence of drug-induced parkinsonism, metabolic identified neurogenetic disorders, encephalitis, or other atypical Parkinsonian syndromes
* Participant with medical history of electroconvulsive therapy or stereotaxic brain surgery for Parkinson's Disease
* Participant with medical history of suicide attempt within 2 years of screening or current suicidal ideation
* Participant with medical history of impulse control disorder

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Sage Investigational Site, Panorama City, California
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Winter Park, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Farmington Hills, Michigan
  - Sage Investigational Site, Berlin, New Jersey
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Orem, Utah

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 9 sites in the United States and took part in the study which ran from 30 November 2016 to 11 September 2017.
Period: Overall Study
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217 | Part B: Antiparkinsonian Agent(s) + SAGE-217
Started | 15 | 14
Completed | 14 | 14
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who were administered study drug [SAGE-217 or levodopa (Part A); or SAGE-217 or antiparkinsonian agent(s) (Part B)].
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217 | Part B: Antiparkinsonian Agent(s) + SAGE-217 | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (6.59) | 65.1 (7.76) | 64.5 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 13 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 14 | 12 | 26
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) - Part A
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. A TEAE was as an AE that occurred after the first administration of study drug. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug (SAGE-217 or levodopa). Overall number of participants analyzed = Number of participants in the safety population that remained in the study during each period.
Measure: Number; unit: percentage of participants
Groups:
- Part A: Antiparkinsonian Agent(s) Day 1 to Day 3: Participants received levodopa as antiparkinsonian agents at the normally prescribed dosing schedule, orally for Days 1 to 3.
- Part A: SAGE-217 Day 4 to Day 7: Participants received SAGE-217 at a dose of 30 mg per day, oral solution, for Days 4 to 7 in the morning with food. If the initial dose was not tolerated, doses could be reduced to 10 or 20 mg per day.
- Part A: Follow-up: Participants resumed levodopa as antiparkinsonian agents at the normally prescribed dosing schedule for Days 8 to 14.
Arm/Group | Part A: Antiparkinsonian Agent(s) Day 1 to Day 3 | Part A: SAGE-217 Day 4 to Day 7 | Part A: Follow-up
Number analyzed (Participants) | 15 | 14 | 15
percentage of participants | 26.7 | 100 | 13.3

2. Primary Outcome: Percentage of Participants With TEAEs, Graded by Severity - Part A
Description: Severity was assessed according to the following scale: mild (awareness of sign or symptom, but easily tolerated); moderate (discomfort sufficient to cause interference with normal activities); severe (incapacitating, with an inability to perform normal activities). The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Antiparkinsonian Agent(s) Day 1 to Day 3 | Part A: SAGE-217 Day 4 to Day 7 | Part A: Follow-up
Number analyzed (Participants) | 15 | 14 | 15
percentage of participants
  Mild | 20.0 | 0 | 6.7
  Moderate | 6.7 | 85.7 | 6.7
  Severe | 0 | 14.3 | 0

3. Primary Outcome: Change From Baseline (CFB) in Basophils - Part A
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, reticulocytes and reticulocytes to erythrocytes ratio. Baseline is the last measurement taken before the first dose of the study drug. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug (SAGE-217 or levodopa). Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9 cells/L)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
10^9 cells per liter (10^9 cells/L)
  Baseline | 0.06 (0.051)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.02 (0.043)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | -0.01 (0.036)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.02 (0.038)
  CFB at Day 14 (Follow-up) | -0.02 (0.041)

4. Primary Outcome: CFB in Basophils to Leukocytes Ratio [Percentage (%)] - Part A
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, reticulocytes and reticulocytes to erythrocytes ratio. Baseline is the last measurement taken before the first dose of the study drug. The analysis was performed in participants included in Part A of the study. The blood cell differential (ratio) data are presented as International System (SI) unit, percentage (%).
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
percentage
  Baseline | 0.8 (0.41)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.1 (0.66)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.3 (0.61)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.0 (0.41)
  CFB at Day 14 (Follow-up) | 0.1 (0.35)

5. Primary Outcome: CFB in Eosinophils - Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
10^9 cells/L
  Baseline | 0.17 (0.098)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.07 (0.083)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.04 (0.051)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.02 (0.073)
  CFB at Day 14 (Follow-up) | 0.00 (0.053)

6. Primary Outcome: CFB in Eosinophils to Leukocytes Ratio (%) - Part A
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, reticulocytes and reticulocytes to erythrocytes ratio. Baseline is the last measurement taken before the first dose of the study drug. The analysis was performed in participants included in Part A of the study. The blood cell differential (ratio) data are presented as SI unit, percentage (%).
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
percentage
  Baseline | 2.9 (1.58)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.7 (1.59)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.3 (0.83)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.0 (0.82)
  CFB at Day 14 (Follow-up) | -0.3 (1.11)

7. Primary Outcome: CFB in Erythrocytes - Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12 cells/L)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
10^12 cells per liter (10^12 cells/L)
  Baseline | 4.63 (0.475)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.01 (0.266)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.04 (0.224)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.02 (0.265)
  CFB at Day 14 (Follow-up) | -0.09 (0.226)

8. Primary Outcome: CFB in Hematocrit - Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters per liter (L/L)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
liters per liter (L/L)
  Baseline | 0.434 (0.0444)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.003 (0.0264)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.004 (0.0247)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | -0.002 (0.0285)
  CFB at Day 14 (Follow-up) | -0.013 (0.0222)

9. Primary Outcome: CFB in Hemoglobin - Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
grams per liter (g/L)
  Baseline | 142.0 (13.87)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.1 (7.55)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 1.7 (7.25)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 1.2 (8.14)
  CFB at Day 14 (Follow-up) | -1.9 (5.82)

10. Primary Outcome: CFB in Leukocytes - Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
10^9 cells/L
  Baseline | 6.04 (1.139)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.24 (1.085)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.15 (0.536)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | -0.09 (0.874)
  CFB at Day 14 (Follow-up) | 0.30 (0.941)

11. Primary Outcome: CFB in Lymphocytes - Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
10^9 cells/L
  Baseline | 1.70 (0.318)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.02 (0.289)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.07 (0.352)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.02 (0.286)
  CFB at Day 14 (Follow-up) | -0.17 (0.183)

12. Primary Outcome: CFB in Lymphocytes to Leukocytes Ratio (%) - Part A
Description: as for outcome 6
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
percentage
  Baseline | 28.3 (4.68)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 1.0 (4.72)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 1.0 (5.55)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.9 (4.87)
  CFB at Day 14 (Follow-up) | -3.9 (4.22)

13. Primary Outcome: CFB in Monocytes - Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
10^9 cells/L
  Baseline | 0.36 (0.112)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.02 (0.125)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.06 (0.076)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.02 (0.101)
  CFB at Day 14 (Follow-up) | 0.05 (0.064)

14. Primary Outcome: CFB in Monocytes to Leukocytes Ratio (%) - Part A
Description: as for outcome 6
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
percentage
  Baseline | 6.1 (1.06)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.2 (1.48)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.6 (1.45)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.5 (1.33)
  CFB at Day 14 (Follow-up) | 0.3 (1.22)

15. Primary Outcome: CFB in Neutrophils- Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
10^9 cells/L
  Baseline | 3.79 (0.861)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.27 (0.848)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | -0.03 (0.599)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | -0.17 (0.680)
  CFB at Day 14 (Follow-up) | 0.44 (0.861)

16. Primary Outcome: CFB in Neutrophils to Leukocytes Ratio (%) - Part A
Description: as for outcome 6
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
percentage
  Baseline | 62.5 (4.26)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -2.4 (4.94)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | -2.4 (5.58)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | -2.2 (4.86)
  CFB at Day 14 (Follow-up) | 3.6 (4.64)

17. Primary Outcome: CFB in Platelets - Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
10^9 cells/L
  Baseline | 218.9 (62.00)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 6.6 (27.07)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 6.8 (33.01)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 7.8 (21.29)
  CFB at Day 14 (Follow-up) | 11.5 (36.42)

18. Primary Outcome: CFB in Reticulocytes - Part A
Description: as for outcome 3
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
10^9 cells/L
  Baseline | 64.6 (20.36)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.3 (17.87)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 12
  CFB at Day 6 (SAGE-217) | 0.3 (19.21)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.2 (20.18)
  CFB at Day 14 (Follow-up) | 0.3 (14.10)

19. Primary Outcome: CFB in Reticulocytes to Erythrocytes Ratio (%) - Part A
Description: as for outcome 6
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
percentage
  Baseline | 1.41 (0.442)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.00 (0.349)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 12
  CFB at Day 6 (SAGE-217) | -0.03 (0.409)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.00 (0.424)
  CFB at Day 14 (Follow-up) | 0.03 (0.315)

20. Primary Outcome: CFB in Activated Partial Thromboplastin Time - Part A
Description: Coagulation measures included activated partial thromboplastin time, prothrombin international normalized ratio and prothrombin time. Baseline is the last measurement taken before the first dose of the study drug. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: seconds (sec)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 13
seconds (sec)
  Baseline | 24.80 [22.9 to 27.4]
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 12
  CFB at Day 4 (SAGE-217) | 0.20 [-1.5 to 4.0]
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 12
  CFB at Day 6 (SAGE-217) | -0.25 [-4.8 to 2.4]
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 11
  CFB at Day 8 (Follow-up) | -0.10 [-1.6 to 1.4]
  CFB at Day 14 (Follow-up) | -1.10 [-2.1 to 4.7]

21. Primary Outcome: CFB in Prothrombin International Normalized Ratio - Part A
Description: as for outcome 20
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 13
ratio
  Baseline | 1.04 (0.065)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 12
  CFB at Day 4 (SAGE-217) | 0.01 (0.108)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 12
  CFB at Day 6 (SAGE-217) | -0.03 (0.065)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 12
  CFB at Day 8 (Follow-up) | 0.05 (0.243)
  CFB at Day 14 (Follow-up) | 0.01 (0.155)

22. Primary Outcome: CFB in Prothrombin Time - Part A
Description: as for outcome 20
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: sec
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 13
sec
  Baseline | 10.70 [10.2 to 12.4]
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 12
  CFB at Day 4 (SAGE-217) | 0.00 [-0.6 to 2.2]
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 12
  CFB at Day 6 (SAGE-217) | 0.00 [-1.2 to 0.4]
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 12
  CFB at Day 8 (Follow-up) | 0.10 [-0.7 to 7.5]
  CFB at Day 14 (Follow-up) | -0.10 [-1.2 to 4.7]

23. Primary Outcome: CFB in Alanine Aminotransferase - Part A
Description: Clinical chemistry measures included alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bicarbonate, bilirubin, calcium, chloride, creatinine, lipase, magnesium, phosphate, potassium, protein, sodium, urate and urea nitrogen. Baseline is the last measurement taken before the first dose of the study drug. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
units per liter (U/L)
  Baseline | 15.8 (8.12)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 15.3 (11.61)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 13.9 (11.87)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 7.2 (13.64)
  CFB at Day 14 (Follow-up) | 2.3 (9.24)

24. Primary Outcome: CFB in Albumin - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
g/L
  Baseline | 43.2 (1.70)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -1.2 (1.81)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | -0.4 (2.59)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -0.1 (2.21)
  CFB at Day 14 (Follow-up) | -0.3 (2.35)

25. Primary Outcome: CFB in Alkaline Phosphatase - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
U/L
  Baseline | 80.6 (14.17)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -1.7 (9.34)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | -2.4 (4.52)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -0.5 (4.78)
  CFB at Day 14 (Follow-up) | 0.0 (8.06)

26. Primary Outcome: CFB in Aspartate Aminotransferase - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
U/L
  Baseline | 23.2 (7.24)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.4 (6.15)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217) | -2.4 (4.93)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -1.0 (5.25)
  CFB at Day 14 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 14 (Follow-up) | 1.8 (5.16)

27. Primary Outcome: CFB in Bicarbonate - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
millimoles per liter (mmol/L)
  Baseline | 22.4 (2.50)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.9 (2.27)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.3 (2.23)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -0.1 (2.41)
  CFB at Day 14 (Follow-up) | 0.7 (2.26)

28. Primary Outcome: CFB in Bilirubin - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micromoles per liter (umol/L)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
micromoles per liter (umol/L)
  Baseline | 6.082 (3.8041)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.029 (3.4758)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.949 (3.8554)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 1.545 (3.5965)
  CFB at Day 14 (Follow-up) | 0.543 (3.7159)

29. Primary Outcome: CFB in Calcium - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmol/L
  Baseline | 2.342 (0.0588)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.030 (0.0734)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.007 (0.0779)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -0.014 (0.0711)
  CFB at Day 14 (Follow-up) | -0.015 (0.0842)

30. Primary Outcome: CFB in Chloride - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmol/L
  Baseline | 100.1 (2.33)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 1.6 (1.91)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 1.1 (2.30)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.5 (2.41)
  CFB at Day 14 (Follow-up) | 0.3 (1.83)

31. Primary Outcome: CFB in Creatinine - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
umol/L
  Baseline | 73.254 (17.7960)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 2.399 (8.6574)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 4.104 (9.4424)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 4.420 (10.9866)
  CFB at Day 14 (Follow-up) | 0.118 (4.6761)

32. Primary Outcome: CFB in Lipase - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
U/L
  Baseline | 34.5 (10.16)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 16.6 (22.15)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 35.1 (77.58)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 73.3 (222.02)
  CFB at Day 14 (Follow-up) | -1.6 (7.67)

33. Primary Outcome: CFB in Magnesium - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmol/L
  Baseline | 0.861 (0.0686)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.012 (0.0409)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.000 (0.0457)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.015 (0.0617)
  CFB at Day 14 (Follow-up) | 0.016 (0.0618)

34. Primary Outcome: CFB in Phosphate - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmol/L
  Baseline | 1.098 (0.1189)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.035 (0.1413)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.076 (0.1645)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.083 (0.1513)
  CFB at Day 14 (Follow-up) | -0.034 (0.1698)

35. Primary Outcome: CFB in Potassium - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmol/L
  Baseline | 4.53 (0.326)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.14 (0.323)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | -0.08 (0.309)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -0.15 (0.350)
  CFB at Day 14 (Follow-up) | -0.08 (0.446)

36. Primary Outcome: CFB in Protein - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
g/L
  Baseline | 69.4 (3.07)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -2.3 (4.12)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | -1.5 (3.86)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -0.4 (3.65)
  CFB at Day 14 (Follow-up) | -1.1 (4.33)

37. Primary Outcome: CFB in Sodium - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmol/L
  Baseline | 140.0 (1.73)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.8 (2.15)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 1.3 (1.86)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.7 (2.20)
  CFB at Day 14 (Follow-up) | 0.5 (1.85)

38. Primary Outcome: CFB in Urate - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmol/L
  Baseline | 0.337 (0.1000)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.005 (0.0713)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.010 (0.0804)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.014 (0.0394)
  CFB at Day 14 (Follow-up) | -0.014 (0.0649)

39. Primary Outcome: CFB in Urea Nitrogen - Part A
Description: as for outcome 23
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmol/L
  Baseline | 5.831 (1.3672)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.587 (1.4925)
  CFB at Day 6 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217) | 0.816 (1.4715)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.663 (1.5521)
  CFB at Day 14 (Follow-up) | -0.048 (1.3484)

40. Primary Outcome: CFB in Specific Gravity - Part A
Description: Urinalysis measures included specific gravity and potential of hydrogen (pH). Baseline is the last measurement taken before the first dose of study drug. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
ratio
  Baseline | 1.018 (0.0049)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | -0.001 (0.0062)
  CFB at Day 7 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217) | 0.000 (0.0039)
  CFB at Day 14 (Follow-up) | 0.002 (0.0059)

41. Primary Outcome: CFB in pH - Part A
Description: Urinalysis measures included specific gravity and pH. Baseline is the last measurement taken before the first dose of study drug. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
pH
  Baseline | 5.87 (0.915)
  CFB at Day 4 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217) | 0.18 (0.973)
  CFB at Day 7 (SAGE-217): number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217) | -0.11 (0.881)
  CFB at Day 14 (Follow-up) | -0.07 (0.884)

42. Primary Outcome: CFB in Temperature - Part A
Description: Vital sign measures included temperature, heart rate, respiratory rate, supine systolic blood pressure, standing systolic blood pressure, supine diastolic blood pressure, standing diastolic blood pressure and pulse oximetry. Baseline is the last measurement taken before the first dose of study drug. L/C indicated levodopa/carbidopa. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees Celsius (degrees C)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
degrees Celsius (degrees C)
  Baseline | 36.61 (0.228)
  CFB at Day 1 (L/C): 1 Hour Postdose | -0.04 (0.180)
  CFB at Day 1 (L/C): 2 Hours Postdose | -0.01 (0.205)
  CFB at Day 1 (L/C): 3 Hours Postdose | -0.05 (0.236)
  CFB at Day 1 (L/C): 4 Hours Postdose | -0.08 (0.227)
  CFB at Day 1 (L/C): 6 Hours Postdose | -0.06 (0.285)
  CFB at Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 8 Hours Postdose | 0.00 (0.235)
  CFB at Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 12 Hours Postdose | 0.08 (0.412)
  CFB at Day 1 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 14 Hours Postdose | 0.00 (0.319)
  CFB at Day 1 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 16 Hours Postdose | -0.01 (0.296)
  CFB at Day 2 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): Predose | -0.06 (0.346)
  CFB at Day 2 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 1 Hour Postdose | -0.11 (0.316)
  CFB at Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 2 Hours Postdose | -0.05 (0.348)
  CFB at Day 2 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 3 Hours Postdose | -0.04 (0.323)
  CFB at Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 4 Hours Postdose | -0.07 (0.279)
  CFB at Day 2 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 6 Hours Postdose | -0.11 (0.274)
  CFB at Day 2 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 8 Hours Postdose | -0.02 (0.283)
  CFB at Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 12 Hours Postdose | 0.06 (0.380)
  CFB at Day 2 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 14 Hours Postdose | -0.05 (0.380)
  CFB at Day 2 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 16 Hours Postdose | -0.06 (0.365)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | 0.09 (0.409)
  CFB at Day 3 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 1 Hour Postdose | -0.09 (0.305)
  CFB at Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 2 Hours Postdose | -0.10 (0.277)
  CFB at Day 3 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 3 Hours Postdose | -0.10 (0.272)
  CFB at Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 4 Hours Postdose | -0.03 (0.331)
  CFB at Day 3 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 6 Hours Postdose | -0.06 (0.363)
  CFB at Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 8 Hours Postdose | -0.04 (0.276)
  CFB at Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 12 Hours Postdose | -0.05 (0.422)
  CFB at Day 3 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 14 Hours Postdose | -0.01 (0.372)
  CFB at Day 3 (L/C): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 16 Hours Postdose | 0.04 (0.176)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 0.02 (0.208)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | 0.01 (0.175)
  CFB at Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 2 Hours Postdose | 0.08 (0.387)
  CFB at Day 4 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 3 Hours Postdose | -0.07 (0.236)
  CFB at Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 4 Hours Postdose | -0.11 (0.236)
  CFB at Day 4 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 6 Hours Postdose | 0.03 (0.230)
  CFB at Day 4 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 8 Hours Postdose | -0.03 (0.336)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | -0.02 (0.333)
  CFB at Day 4 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 14 Hours Postdose | 0.12 (0.185)
  CFB at Day 4 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 16 Hours Postdose | 0.07 (0.233)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | -0.05 (0.187)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -0.04 (0.287)
  CFB at Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 12
  CFB at Day 5 (SAGE-217): 2 Hours Postdose | -0.16 (0.360)
  CFB at Day 5 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 3 Hours Postdose | -0.17 (0.272)
  CFB at Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 4 Hours Postdose | -0.02 (0.449)
  CFB at Day 5 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 6 Hours Postdose | -0.16 (0.310)
  CFB at Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 8 Hours Postdose | -0.07 (0.421)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | -0.09 (0.400)
  CFB at Day 5 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 14 Hours Postdose | -0.07 (0.273)
  CFB at Day 5 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 16 Hours Postdose | -0.02 (0.383)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -0.04 (0.359)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | 0.02 (0.306)
  CFB at Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 2 Hours Postdose | -0.08 (0.322)
  CFB at Day 6 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 3 Hours Postdose | -0.13 (0.322)
  CFB at Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 4 Hours Postdose | -0.12 (0.358)
  CFB at Day 6 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 6 Hours Postdose | -0.09 (0.260)
  CFB at Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 8 Hours Postdose | -0.08 (0.329)
  CFB at Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 12 Hours Postdose | -0.10 (0.697)
  CFB at Day 6 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 14 Hours Postdose | -0.04 (0.434)
  CFB at Day 6 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 16 Hours Postdose | 0.06 (0.434)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | -0.13 (0.302)
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | -0.16 (0.282)
  CFB at Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 2 Hours Postdose | -0.16 (0.407)
  CFB at Day 7 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 3 Hours Postdose | -0.16 (0.310)
  CFB at Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 4 Hours Postdose | -0.11 (0.332)
  CFB at Day 7 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 6 Hours Postdose | -0.13 (0.252)
  CFB at Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 8 Hours Postdose | 0.02 (0.208)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | 0.06 (0.145)
  CFB at Day 7 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 14 Hours Postdose | -0.01 (0.235)
  CFB at Day 7 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 16 Hours Postdose | -0.03 (0.363)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.4 (0.224)
  CFB at Day 14 (Follow-up) | 0.07 (0.301)

43. Primary Outcome: CFB in Heart Rate - Part A
Description: as for outcome 42
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
beats per minute (beats/min)
  Baseline | 66.6 (11.83)
  CFB at Day 1 (L/C): 1 Hour Postdose | 2.1 (5.87)
  CFB at Day 1 (L/C): 2 Hours Postdose | 1.3 (6.76)
  CFB at Day 1 (L/C): 3 Hours Postdose | -0.5 (5.87)
  CFB at Day 1 (L/C): 4 Hours Postdose | -1.3 (6.63)
  CFB at Day 1 (L/C): 6 Hours Postdose | 0.8 (7.75)
  CFB at Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 8 Hours Postdose | 0.4 (7.55)
  CFB at Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 12 Hours Postdose | 5.5 (6.86)
  CFB at Day 1 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 14 Hours Postdose | 0.5 (7.18)
  CFB at Day 1 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 16 Hours Postdose | 1.4 (5.03)
  CFB at Day 2 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): Predose | -0.2 (6.80)
  CFB at Day 2 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 1 Hour Postdose | 2.1 (7.37)
  CFB at Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 2 Hours Postdose | 1.9 (8.10)
  CFB at Day 2 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 3 Hours Postdose | -0.3 (10.71)
  CFB at Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 4 Hours Postdose | -0.9 (5.23)
  CFB at Day 2 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 6 Hours Postdose | 2.1 (7.08)
  CFB at Day 2 (L/C): 8 Hours Postdos: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 8 Hours Postdos | 3.8 (7.81)
  CFB at Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 12 Hours Postdose | 3.9 (8.38)
  CFB at Day 2 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 14 Hours Postdose | 1.6 (7.29)
  CFB at Day 2 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 16 Hours Postdose | 1.2 (7.29)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -0.7 (9.29)
  CFB at Day 3 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 1 Hour Postdose | 4.7 (6.67)
  CFB at Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 2 Hours Postdose | 2.4 (9.46)
  CFB at Day 3 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 3 Hours Postdose | 1.2 (7.20)
  CFB at Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 4 Hours Postdose | 0.6 (6.30)
  CFB at Day 3 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 6 Hours Postdose | 1.7 (7.33)
  CFB at Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 8 Hours Postdose | 5.9 (5.43)
  CFB at Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 12 Hours Postdose | 2.6 (9.72)
  CFB at Day 3 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 14 Hours Postdose | 3.6 (8.63)
  CFB at Day 3 (L/C): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 16 Hours Postdose | 3.9 (7.08)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 1.4 (5.21)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | 3.7 (6.43)
  CFB at Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 2 Hours Postdose | 1.6 (8.97)
  CFB at Day 4 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 3 Hours Postdose | 3.4 (10.38)
  CFB at Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 4 Hours Postdose | 0.6 (6.27)
  CFB at Day 4 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 6 Hours Postdose | 2.7 (8.72)
  CFB at Day 4 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 8 Hours Postdose | 2.1 (7.97)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 5.1 (9.70)
  CFB at Day 4 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 14 Hours Postdose | 5.2 (6.64)
  CFB at Day 4 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 16 Hours Postdose | 4.6 (7.37)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | 1.5 (8.25)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | 3.8 (6.99)
  CFB at Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 2 Hours Postdose | 4.4 (9.06)
  CFB at Day 5 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 3 Hours Postdose | 3.4 (8.18)
  CFB at Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 4 Hours Postdose | 1.3 (11.03)
  CFB at Day 5 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 6 Hours Postdose | 7.6 (11.24)
  CFB at Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 8 Hours Postdose | 4.2 (9.50)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | 8.4 (9.51)
  CFB at Day 5 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 14 Hours Postdose | 6.6 (7.98)
  CFB at Day 5 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 16 Hours Postdose | 3.7 (9.34)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | 4.6 (7.58)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | 4.3 (6.53)
  CFB at Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 2 Hours Postdose | 2.9 (7.86)
  CFB at Day 6 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 3 Hours Postdose | 4.2 (7.51)
  CFB at Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 4 Hours Postdose | 3.2 (10.09)
  CFB at Day 6 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 6 Hours Postdose | 5.1 (10.07)
  CFB at Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 8 Hours Postdose | 4.6 (11.00)
  CFB at Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 12 Hours Postdose | 4.8 (10.87)
  CFB at Day 6 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 14 Hours Postdose | 5.2 (9.51)
  CFB at Day 6 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 16 Hours Postdose | 5.4 (10.87)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | 8.4 (11.06)
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | 6.0 (8.29)
  CFB at Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 2 Hours Postdose | 5.3 (6.49)
  CFB at Day 7 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 3 Hours Postdose | 3.9 (12.50)
  CFB at Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 4 Hours Postdose | 4.4 (7.77)
  CFB at Day 7 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 6 Hours Postdose | 6.0 (8.46)
  CFB at Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 8 Hours Postdose | 4.8 (4.66)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | 9.5 (9.82)
  CFB at Day 7 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 14 Hours Postdose | 6.7 (9.27)
  CFB at Day 7 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 16 Hours Postdose | 5.6 (7.93)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 1.8 (6.52)
  CFB at Day 14 (Follow-up) | 4.1 (8.29)

44. Primary Outcome: CFB in Respiratory Rate - Part A
Description: as for outcome 42
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: breaths per minute (breaths/min)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
breaths per minute (breaths/min)
  Baseline | 15.9 (1.92)
  CFB at Day 1 (L/C): 1 Hour Postdose | 0.1 (1.46)
  CFB at Day 1 (L/C): 2 Hours Postdose | 0.1 (1.92)
  CFB at Day 1 (L/C): 3 Hours Postdose | 0.0 (1.69)
  CFB at Day 1 (L/C): 4 Hours Postdose | 0.2 (1.93)
  CFB at Day 1 (L/C): 6 Hours Postdose | 0.0 (1.69)
  CFB at Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 8 Hours Postdose | 1.0 (2.08)
  CFB at Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 12 Hours Postdose | 0.6 (1.99)
  CFB at Day 1 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 14 Hours Postdose | 0.1 (1.83)
  CFB at Day 1 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 16 Hours Postdose | -0.2 (2.49)
  CFB at Day 2 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): Predose | -0.1 (1.59)
  CFB at Day 2 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 1 Hour Postdose | 0.1 (1.83)
  CFB at Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 2 Hours Postdose | 0.2 (1.48)
  CFB at Day 2 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 3 Hours Postdose | 0.0 (1.57)
  CFB at Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 4 Hours Postdose | 0.5 (1.70)
  CFB at Day 2 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 6 Hours Postdose | 0.4 (2.14)
  CFB at Day 2 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 8 Hours Postdose | 0.1 (2.32)
  CFB at Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 12 Hours Postdose | 0.3 (2.61)
  CFB at Day 2 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 14 Hours Postdose | 0.3 (2.92)
  CFB at Day 2 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 16 Hours Postdose | 0.1 (2.62)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -0.4 (1.99)
  CFB at Day 3 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 1 Hour Postdose | 0.4 (1.65)
  CFB at Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 2 Hours Postdose | -0.1 (2.03)
  CFB at Day 3 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 3 Hours Postdose | 0.4 (2.13)
  CFB at Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 4 Hours Postdose | 0.1 (2.11)
  CFB at Day 3 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 6 Hours Postdose | 0.4 (1.87)
  CFB at Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 8 Hours Postdose | 0.2 (2.26)
  CFB at Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 12 Hours Postdose | 0.4 (1.65)
  CFB at Day 3 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 14 Hours Postdose | 0.2 (1.93)
  CFB at Day 3 (L/C): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 16 Hours Postdose | 0.0 (2.74)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 0.9 (1.59)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | -0.3 (2.69)
  CFB at Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 2 Hours Postdose | -0.4 (2.79)
  CFB at Day 4 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 3 Hours Postdose | 0.3 (2.39)
  CFB at Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 4 Hours Postdose | -0.1 (1.66)
  CFB at Day 4 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 6 Hours Postdose | 0.1 (1.21)
  CFB at Day 4 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 8 Hours Postdose | 0.7 (1.68)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 0.9 (1.86)
  CFB at Day 4 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 14 Hours Postdose | 0.5 (1.70)
  CFB at Day 4 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 16 Hours Postdose | -0.3 (2.02)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | -0.1 (1.59)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -0.3 (2.20)
  CFB at Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 2 Hours Postdose | -0.4 (2.34)
  CFB at Day 5 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 3 Hours Postdose | -0.1 (1.77)
  CFB at Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 4 Hours Postdose | 0.1 (1.86)
  CFB at Day 5 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 6 Hours Postdose | 0.4 (2.27)
  CFB at Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 8 Hours Postdose | 1.0 (1.92)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | 0.4 (1.95)
  CFB at Day 5 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 14 Hours Postdose | 0.5 (1.95)
  CFB at Day 5 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 16 Hours Postdose | 0.3 (2.05)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -0.1 (1.38)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | -0.6 (1.65)
  CFB at Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 2 Hours Postdose | -0.3 (1.38)
  CFB at Day 6 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 3 Hours Postdose | -0.1 (2.18)
  CFB at Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 4 Hours Postdose | -0.1 (1.79)
  CFB at Day 6 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 6 Hours Postdose | 0.4 (2.21)
  CFB at Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 8 Hours Postdose | 1.0 (1.92)
  CFB at Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 12 Hours Postdose | 0.4 (2.82)
  CFB at Day 6 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 14 Hours Postdose | 0.5 (2.10)
  CFB at Day 6 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 16 Hours Postdose | 0.4 (2.31)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | 0.0 (1.36)
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | 0.1 (1.27)
  CFB at Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 2 Hours Postdose | 0.9 (1.51)
  CFB at Day 7 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 3 Hours Postdose | 0.1 (1.49)
  CFB at Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 4 Hours Postdose | 0.1 (1.66)
  CFB at Day 7 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 6 Hours Postdose | 0.6 (1.65)
  CFB at Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 8 Hours Postdose | 0.4 (1.65)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | 1.4 (2.03)
  CFB at Day 7 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 14 Hours Postdose | 0.4 (2.31)
  CFB at Day 7 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 16 Hours Postdose | 0.7 (2.61)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.1 (1.29)
  CFB at Day 14 (Follow-up) | 0.9 (1.83)

45. Primary Outcome: CFB in Supine Systolic Blood Pressure - Part A
Description: as for outcome 42
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
millimeters of mercury (mmHg)
  Baseline | 124.5 (11.61)
  CFB at Day 1 (L/C): 1 Hour Postdose | -6.7 (10.81)
  CFB at Day 1 (L/C): 2 Hours Postdose | -7.1 (11.49)
  CFB at Day 1 (L/C): 3 Hours Postdose | -1.5 (10.37)
  CFB at Day 1 (L/C): 4 Hours Postdose | -4.7 (9.44)
  CFB at Day 1 (L/C): 6 Hours Postdose | -4.5 (9.63)
  CFB at Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 8 Hours Postdose | 2.4 (13.32)
  CFB at Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 12 Hours Postdose | 3.4 (13.21)
  CFB at Day 1 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 14 Hours Postdose | -3.0 (12.51)
  CFB at Day 1 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 16 Hours Postdose | -3.9 (11.99)
  CFB at Day 2 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): Predose | -0.4 (11.14)
  CFB at Day 2 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 1 Hour Postdose | -7.3 (11.59)
  CFB at Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 2 Hours Postdose | -4.4 (9.99)
  CFB at Day 2 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 3 Hours Postdose | -0.8 (10.86)
  CFB at Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 4 Hours Postdose | -1.1 (10.43)
  CFB at Day 2 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 6 Hours Postdose | -1.6 (10.95)
  CFB at Day 2 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 8 Hours Postdose | 3.2 (15.35)
  CFB at Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 12 Hours Postdose | 5.9 (8.00)
  CFB at Day 2 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 14 Hours Postdose | 3.4 (9.53)
  CFB at Day 2 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 16 Hours Postdose | 0.9 (10.40)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | 1.2 (8.61)
  CFB at Day 3 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 1 Hour Postdose | -2.5 (10.30)
  CFB at Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 2 Hours Postdose | -7.4 (14.70)
  CFB at Day 3 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 3 Hours Postdose | -3.1 (12.69)
  CFB at Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 4 Hours Postdose | -3.7 (14.12)
  CFB at Day 3 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 6 Hours Postdose | -3.1 (12.51)
  CFB at Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 8 Hours Postdose | -1.3 (12.75)
  CFB at Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 12 Hours Postdose | 3.3 (13.30)
  CFB at Day 3 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 14 Hours Postdose | 3.6 (16.21)
  CFB at Day 3 (L/C): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 16 Hours Postdose | -3.3 (10.73)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 3.5 (10.17)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | -4.8 (9.75)
  CFB at Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 2 Hours Postdose | -6.6 (10.80)
  CFB at Day 4 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 3 Hours Postdose | 2.3 (15.97)
  CFB at Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 4 Hours Postdose | -1.6 (8.84)
  CFB at Day 4 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 6 Hours Postdose | -3.9 (10.46)
  CFB at Day 4 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 8 Hours Postdose | 2.2 (10.94)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 3.1 (9.60)
  CFB at Day 4 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 14 Hours Postdose | -3.1 (14.15)
  CFB at Day 4 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 16 Hours Postdose | -2.6 (10.83)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | 0.1 (11.43)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -8.6 (9.68)
  CFB at Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 2 Hours Postdose | -8.1 (11.67)
  CFB at Day 5 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 3 Hours Postdose | -5.8 (10.14)
  CFB at Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 4 Hours Postdose | -0.4 (9.23)
  CFB at Day 5 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 6 Hours Postdose | -2.9 (11.14)
  CFB at Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 8 Hours Postdose | -3.8 (10.15)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | 1.3 (11.68)
  CFB at Day 5 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 14 Hours Postdose | 1.7 (15.46)
  CFB at Day 5 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 16 Hours Postdose | 0.6 (14.19)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -5.9 (11.67)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | -8.6 (11.95)
  CFB at Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 2 Hours Postdose | -3.8 (13.03)
  CFB at Day 6 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 3 Hours Postdose | -4.1 (15.47)
  CFB at Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 4 Hours Postdose | -5.6 (13.00)
  CFB at Day 6 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 6 Hours Postdose | -4.4 (10.23)
  CFB at Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 8 Hours Postdose | -0.1 (12.46)
  CFB at Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 12 Hours Postdose | -0.1 (12.41)
  CFB at Day 6 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 14 Hours Postdose | 2.5 (10.39)
  CFB at Day 6 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 16 Hours Postdose | 1.8 (13.45)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | 1.9 (19.64)
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | -5.9 (12.93)
  CFB at Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 2 Hours Postdose | -5.4 (18.93)
  CFB at Day 7 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 3 Hours Postdose | -2.8 (13.22)
  CFB at Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 4 Hours Postdose | -5.1 (17.35)
  CFB at Day 7 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 6 Hours Postdose | -3.9 (14.81)
  CFB at Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 8 Hours Postdose | -3.1 (10.38)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | 2.9 (13.23)
  CFB at Day 7 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 14 Hours Postdose | -0.6 (14.07)
  CFB at Day 7 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 16 Hours Postdose | -0.2 (18.75)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 1.7 (7.79)
  CFB at Day 14 (Follow-up) | 2.7 (9.50)

46. Primary Outcome: CFB in Standing Systolic Blood Pressure - Part A
Description: as for outcome 42
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmHg
  Baseline | 124.1 (12.38)
  CFB at Day 1 (L/C): 1 Hour Postdose | -3.1 (9.98)
  CFB at Day 1 (L/C): 2 Hours Postdose | -4.7 (10.00)
  CFB at Day 1 (L/C): 3 Hours Postdose | -2.9 (11.45)
  CFB at Day 1 (L/C): 4 Hours Postdose | 0.0 (11.78)
  CFB at Day 1 (L/C): 6 Hours Postdose | 2.7 (13.34)
  CFB at Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 8 Hours Postdose | 4.3 (10.22)
  CFB at Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 12 Hours Postdose | 7.6 (17.85)
  CFB at Day 1 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 14 Hours Postdose | 2.9 (10.18)
  CFB at Day 1 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 16 Hours Postdose | -2.7 (9.51)
  CFB at Day 2 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): Predose | 1.0 (11.09)
  CFB at Day 2 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 1 Hour Postdose | -2.9 (10.57)
  CFB at Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 2 Hours Postdose | -3.4 (11.56)
  CFB at Day 2 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 3 Hours Postdose | -5.1 (9.86)
  CFB at Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 4 Hours Postdose | 0.0 (10.12)
  CFB at Day 2 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 6 Hours Postdose | -3.4 (8.50)
  CFB at Day 2 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 8 Hours Postdose | -0.6 (10.20)
  CFB at Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 12 Hours Postdose | 5.6 (16.97)
  CFB at Day 2 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 14 Hours Postdose | 2.0 (11.08)
  CFB at Day 2 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 16 Hours Postdose | -4.4 (10.14)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -1.4 (7.84)
  CFB at Day 3 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 1 Hour Postdose | -4.2 (8.17)
  CFB at Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 2 Hours Postdose | -4.9 (11.83)
  CFB at Day 3 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 3 Hours Postdose | -4.4 (13.07)
  CFB at Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 4 Hours Postdose | -6.2 (13.13)
  CFB at Day 3 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 6 Hours Postdose | -3.2 (9.35)
  CFB at Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 8 Hours Postdose | -3.2 (10.83)
  CFB at Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 12 Hours Postdose | 1.8 (14.56)
  CFB at Day 3 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 14 Hours Postdose | 0.0 (15.65)
  CFB at Day 3 (L/C): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 16 Hours Postdose | 2.2 (11.98)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 3.3 (13.32)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 10
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | -1.5 (14.74)
  CFB at Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 11
  CFB at Day 4 (SAGE-217): 2 Hours Postdose | -4.6 (10.60)
  CFB at Day 4 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 3 Hours Postdose | -0.5 (11.77)
  CFB at Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 4 Hours Postdose | -5.7 (10.04)
  CFB at Day 4 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 6 Hours Postdose | -2.3 (8.50)
  CFB at Day 4 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 8 Hours Postdose | 0.9 (9.16)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 3.3 (12.72)
  CFB at Day 4 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 14 Hours Postdose | 0.0 (10.09)
  CFB at Day 4 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 16 Hours Postdose | -1.3 (10.07)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | -0.6 (9.61)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 11
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -9.8 (12.60)
  CFB at Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 12
  CFB at Day 5 (SAGE-217): 2 Hours Postdose | -8.3 (10.52)
  CFB at Day 5 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 3 Hours Postdose | -3.8 (14.81)
  CFB at Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 4 Hours Postdose | -2.4 (9.82)
  CFB at Day 5 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 6 Hours Postdose | -2.1 (12.05)
  CFB at Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 8 Hours Postdose | -3.3 (10.16)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | 1.4 (12.51)
  CFB at Day 5 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 14 Hours Postdose | 2.3 (17.97)
  CFB at Day 5 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 16 Hours Postdose | 0.8 (15.37)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -3.3 (12.00)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | -6.4 (10.89)
  CFB at Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 2 Hours Postdose | -5.5 (9.34)
  CFB at Day 6 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 3 Hours Postdose | -3.5 (10.36)
  CFB at Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 4 Hours Postdose | -2.8 (8.55)
  CFB at Day 6 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 6 Hours Postdose | 1.6 (9.45)
  CFB at Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 8 Hours Postdose | -2.7 (12.79)
  CFB at Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 12 Hours Postdose | -2.9 (12.13)
  CFB at Day 6 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 14 Hours Postdose | 2.5 (13.57)
  CFB at Day 6 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 16 Hours Postdose | 0.6 (19.21)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | -0.2 (12.25)
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | -4.0 (13.06)
  CFB at Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 2 Hours Postdose | -4.7 (13.19)
  CFB at Day 7 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 3 Hours Postdose | -6.0 (9.27)
  CFB at Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 4 Hours Postdose | -5.9 (13.96)
  CFB at Day 7 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 6 Hours Postdose | -2.4 (13.65)
  CFB at Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 8 Hours Postdose | 2.1 (10.80)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | 4.6 (14.54)
  CFB at Day 7 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 14 Hours Postdose | 3.7 (13.23)
  CFB at Day 7 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 16 Hours Postdose | 0.5 (11.95)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 7.6 (9.90)
  CFB at Day 14 (Follow-up) | 3.6 (13.14)

47. Primary Outcome: CFB in Supine Diastolic Blood Pressure - Part A
Description: as for outcome 42
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmHg
  Baseline | 77.3 (7.19)
  CFB at Day 1 (L/C): 1 Hour Postdose | -5.3 (6.02)
  CFB at Day 1 (L/C): 2 Hours Postdose | -4.7 (5.92)
  CFB at Day 1 (L/C): 3 Hours Postdose | -3.2 (6.66)
  CFB at Day 1 (L/C): 4 Hours Postdose | -3.1 (5.26)
  CFB at Day 1 (L/C): 6 Hours Postdose | -3.9 (9.91)
  CFB at Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 8 Hours Postdose | -0.4 (9.04)
  CFB at Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 12 Hours Postdose | -0.1 (7.89)
  CFB at Day 1 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 14 Hours Postdose | -3.6 (8.94)
  CFB at Day 1 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 16 Hours Postdose | -5.0 (10.34)
  CFB at Day 2 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): Predose | 0.7 (7.10)
  CFB at Day 2 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 1 Hour Postdose | -4.8 (9.49)
  CFB at Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 2 Hours Postdose | -3.4 (9.90)
  CFB at Day 2 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 3 Hours Postdose | -2.2 (11.37)
  CFB at Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 4 Hours Postdose | -2.5 (7.78)
  CFB at Day 2 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 6 Hours Postdose | -1.4 (10.09)
  CFB at Day 2 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 8 Hours Postdose | -1.4 (10.47)
  CFB at Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 12 Hours Postdose | 0.9 (7.57)
  CFB at Day 2 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 14 Hours Postdose | -1.9 (8.08)
  CFB at Day 2 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 16 Hours Postdose | -3.4 (7.13)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -0.8 (7.29)
  CFB at Day 3 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 1 Hour Postdose | -5.1 (8.51)
  CFB at Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 2 Hours Postdose | -3.1 (8.11)
  CFB at Day 3 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 3 Hours Postdose | -4.3 (9.77)
  CFB at Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 4 Hours Postdose | -5.9 (13.63)
  CFB at Day 3 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 6 Hours Postdose | -4.1 (8.77)
  CFB at Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 8 Hours Postdose | -3.9 (9.90)
  CFB at Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 12 Hours Postdose | -1.0 (8.32)
  CFB at Day 3 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 14 Hours Postdose | -0.9 (7.80)
  CFB at Day 3 (L/C): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 16 Hours Postdose | -2.5 (8.69)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 1.8 (7.82)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | -1.9 (6.72)
  CFB at Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 2 Hours Postdose | -3.6 (6.48)
  CFB at Day 4 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 3 Hours Postdose | 1.5 (8.19)
  CFB at Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 4 Hours Postdose | -0.8 (8.01)
  CFB at Day 4 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 6 Hours Postdose | -3.6 (8.75)
  CFB at Day 4 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 8 Hours Postdose | -1.7 (7.08)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 0.0 (6.93)
  CFB at Day 4 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 14 Hours Postdose | -3.6 (8.84)
  CFB at Day 4 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 16 Hours Postdose | -4.0 (7.05)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | -2.1 (8.43)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -5.4 (7.72)
  CFB at Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 2 Hours Postdose | -2.4 (6.17)
  CFB at Day 5 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 3 Hours Postdose | -3.1 (6.62)
  CFB at Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 4 Hours Postdose | -3.3 (6.93)
  CFB at Day 5 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 6 Hours Postdose | -2.4 (8.22)
  CFB at Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 8 Hours Postdose | -3.4 (7.00)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | -4.0 (9.17)
  CFB at Day 5 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 14 Hours Postdose | -4.3 (7.84)
  CFB at Day 5 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 16 Hours Postdose | -2.2 (10.02)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -3.6 (7.59)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | -3.7 (9.72)
  CFB at Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 2 Hours Postdose | -2.7 (9.31)
  CFB at Day 6 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 3 Hours Postdose | -1.8 (8.99)
  CFB at Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 4 Hours Postdose | -1.8 (11.37)
  CFB at Day 6 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 6 Hours Postdose | -3.9 (8.09)
  CFB at Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 8 Hours Postdose | -1.7 (8.06)
  CFB at Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 12 Hours Postdose | -1.0 (9.17)
  CFB at Day 6 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 14 Hours Postdose | 0.8 (7.71)
  CFB at Day 6 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 16 Hours Postdose | -3.6 (10.30)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | -1.9 (6.75)
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | -5.1 (7.79)
  CFB at Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 2 Hours Postdose | -3.5 (9.61)
  CFB at Day 7 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 3 Hours Postdose | -2.7 (10.46)
  CFB at Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 4 Hours Postdose | -4.5 (9.40)
  CFB at Day 7 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 6 Hours Postdose | -4.8 (8.58)
  CFB at Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 8 Hours Postdose | -2.2 (10.02)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | -1.0 (8.58)
  CFB at Day 7 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 14 Hours Postdose | -3.5 (10.65)
  CFB at Day 7 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 16 Hours Postdose | -4.2 (9.66)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -3.8 (8.05)
  CFB at Day 14 (Follow-up) | -2.2 (7.22)

48. Primary Outcome: CFB in Standing Diastolic Blood Pressure - Part A
Description: as for outcome 42
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
mmHg
  Baseline | 76.7 (10.57)
  CFB at Day 1 (L/C): 1 Hour Postdose | 0.4 (8.71)
  CFB at Day 1 (L/C): 2 Hours Postdose | -2.9 (7.26)
  CFB at Day 1 (L/C): 3 Hours Postdose | 0.7 (7.92)
  CFB at Day 1 (L/C): 4 Hours Postdose | 2.3 (5.57)
  CFB at Day 1 (L/C): 6 Hours Postdose | 0.9 (10.54)
  CFB at Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 8 Hours Postdose | 3.1 (7.16)
  CFB at Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 12 Hours Postdose | 2.6 (7.04)
  CFB at Day 1 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 14 Hours Postdose | 1.3 (7.65)
  CFB at Day 1 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 16 Hours Postdose | 1.6 (7.19)
  CFB at Day 2 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): Predose | 4.0 (8.41)
  CFB at Day 2 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 1 Hour Postdose | 1.6 (7.89)
  CFB at Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 2 Hours Postdose | 1.1 (12.25)
  CFB at Day 2 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 3 Hours Postdose | 1.1 (8.53)
  CFB at Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 4 Hours Postdose | 3.8 (10.08)
  CFB at Day 2 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 6 Hours Postdose | 0.3 (12.55)
  CFB at Day 2 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 8 Hours Postdose | 1.6 (10.91)
  CFB at Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 12 Hours Postdose | 4.3 (6.80)
  CFB at Day 2 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 14 Hours Postdose | 3.7 (5.99)
  CFB at Day 2 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 16 Hours Postdose | 0.1 (5.34)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | 4.4 (7.82)
  CFB at Day 3 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 1 Hour Postdose | -1.1 (9.44)
  CFB at Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 2 Hours Postdose | -0.9 (6.98)
  CFB at Day 3 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 3 Hours Postdose | -1.7 (12.74)
  CFB at Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 4 Hours Postdose | -0.7 (11.23)
  CFB at Day 3 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 6 Hours Postdose | -0.6 (9.94)
  CFB at Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 8 Hours Postdose | -1.0 (11.90)
  CFB at Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 12 Hours Postdose | 0.6 (7.43)
  CFB at Day 3 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 14 Hours Postdose | 1.8 (9.57)
  CFB at Day 3 (L/C): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 16 Hours Postdose | 3.8 (10.98)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 4.6 (9.11)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 10
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | 1.8 (8.09)
  CFB at Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 11
  CFB at Day 4 (SAGE-217): 2 Hours Postdose | 2.4 (6.86)
  CFB at Day 4 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 3 Hours Postdose | 5.6 (7.50)
  CFB at Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 4 Hours Postdose | 3.7 (7.90)
  CFB at Day 4 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 6 Hours Postdose | 0.3 (8.17)
  CFB at Day 4 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 8 Hours Postdose | 1.9 (7.88)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 4.8 (11.13)
  CFB at Day 4 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 14 Hours Postdose | 1.9 (10.41)
  CFB at Day 4 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 16 Hours Postdose | 2.8 (9.24)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | 2.6 (5.84)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 11
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -2.5 (5.99)
  CFB at Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 12
  CFB at Day 5 (SAGE-217): 2 Hours Postdose | -0.8 (6.66)
  CFB at Day 5 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 3 Hours Postdose | 3.8 (6.44)
  CFB at Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 4 Hours Postdose | 2.7 (6.34)
  CFB at Day 5 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 6 Hours Postdose | 1.6 (6.21)
  CFB at Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 8 Hours Postdose | 0.1 (8.02)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | 0.2 (9.27)
  CFB at Day 5 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 14 Hours Postdose | 0.4 (9.18)
  CFB at Day 5 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 16 Hours Postdose | 0.8 (9.71)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -0.4 (8.56)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | 0.9 (7.45)
  CFB at Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 2 Hours Postdose | 0.8 (7.10)
  CFB at Day 6 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 3 Hours Postdose | 2.0 (10.43)
  CFB at Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 4 Hours Postdose | 1.2 (8.84)
  CFB at Day 6 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 6 Hours Postdose | 1.6 (7.06)
  CFB at Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 8 Hours Postdose | 2.3 (9.25)
  CFB at Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 12 Hours Postdose | 0.7 (9.63)
  CFB at Day 6 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 14 Hours Postdose | 3.1 (8.10)
  CFB at Day 6 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 16 Hours Postdose | 2.8 (11.44)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | 2.4 (8.24)
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | 0.3 (8.72)
  CFB at Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 2 Hours Postdose | -2.0 (7.54)
  CFB at Day 7 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 3 Hours Postdose | -0.2 (6.47)
  CFB at Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 4 Hours Postdose | -1.4 (9.98)
  CFB at Day 7 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 6 Hours Postdose | -0.9 (7.85)
  CFB at Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 8 Hours Postdose | 2.7 (6.91)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | 2.0 (10.58)
  CFB at Day 7 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 14 Hours Postdose | 2.9 (11.34)
  CFB at Day 7 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 16 Hours Postdose | 1.1 (9.31)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 2.1 (7.47)
  CFB at Day 14 (Follow-up) | 1.5 (8.06)

49. Primary Outcome: CFB in Pulse Oximetry- Part A
Description: as for outcome 42
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
percentage
  Baseline | 96.9 (2.22)
  CFB at Day 1 (L/C): 1 Hour Postdose | -0.3 (1.03)
  CFB at Day 1 (L/C): 2 Hours Postdose | 0.2 (1.42)
  CFB at Day 1 (L/C): 3 Hours Postdose | 0.2 (1.90)
  CFB at Day 1 (L/C): 4 Hours Postdose | 0.1 (2.02)
  CFB at Day 1 (L/C): 6 Hours Postdose | -0.2 (1.42)
  CFB at Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 8 Hours Postdose | -0.1 (1.23)
  CFB at Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 12 Hours Postdose | -0.1 (1.46)
  CFB at Day 1 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 14 Hours Postdose | -0.4 (1.08)
  CFB at Day 1 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 16 Hours Postdose | -0.7 (2.64)
  CFB at Day 2 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): Predose | -0.6 (1.50)
  CFB at Day 2 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 1 Hour Postdose | -0.4 (2.02)
  CFB at Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 2 Hours Postdose | -0.4 (1.83)
  CFB at Day 2 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 3 Hours Postdose | -0.2 (0.97)
  CFB at Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 4 Hours Postdose | -0.7 (2.02)
  CFB at Day 2 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 6 Hours Postdose | -0.5 (2.38)
  CFB at Day 2 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 8 Hours Postdose | 0.4 (1.91)
  CFB at Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 12 Hours Postdose | -0.1 (1.17)
  CFB at Day 2 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 14 Hours Postdose | -0.6 (1.28)
  CFB at Day 2 (L/C): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 16 Hours Postdose | -0.2 (1.31)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -0.5 (1.79)
  CFB at Day 3 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 1 Hour Postdose | -1.1 (1.86)
  CFB at Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 2 Hours Postdose | -0.4 (1.70)
  CFB at Day 3 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 3 Hours Postdose | -0.3 (1.44)
  CFB at Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 4 Hours Postdose | -0.1 (1.33)
  CFB at Day 3 (L/C): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 6 Hours Postdose | 0.3 (1.59)
  CFB at Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 8 Hours Postdose | -0.1 (1.90)
  CFB at Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 12 Hours Postdose | 0.0 (1.36)
  CFB at Day 3 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 14 Hours Postdose | 0.4 (1.28)
  CFB at Day 3 (L/C): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 16 Hours Postdose | -0.2 (1.63)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 0.0 (0.96)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | -1.6 (3.69)
  CFB at Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 2 Hours Postdose | -0.7 (2.73)
  CFB at Day 4 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 3 Hours Postdose | -0.1 (1.82)
  CFB at Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 4 Hours Postdose | -0.4 (1.09)
  CFB at Day 4 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 6 Hours Postdose | -0.4 (1.87)
  CFB at Day 4 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 8 Hours Postdose | -0.4 (1.28)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | -0.1 (1.29)
  CFB at Day 4 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 14 Hours Postdose | -0.2 (1.42)
  CFB at Day 4 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 16 Hours Postdose | -0.3 (1.68)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | 0.2 (1.76)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -1.3 (2.61)
  CFB at Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 2 Hours Postdose | -1.2 (2.72)
  CFB at Day 5 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 3 Hours Postdose | 0.1 (1.82)
  CFB at Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 4 Hours Postdose | 0.0 (1.36)
  CFB at Day 5 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 6 Hours Postdose | -0.2 (1.72)
  CFB at Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 8 Hours Postdose | -0.1 (1.73)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | -0.4 (2.56)
  CFB at Day 5 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 14 Hours Postdose | -0.6 (2.34)
  CFB at Day 5 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 16 Hours Postdose | -1.1 (2.87)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -0.5 (1.61)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | -1.1 (1.59)
  CFB at Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 2 Hours Postdose | 0.1 (2.37)
  CFB at Day 6 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 3 Hours Postdose | -0.9 (2.03)
  CFB at Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 4 Hours Postdose | -0.4 (2.34)
  CFB at Day 6 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 6 Hours Postdose | 0.1 (2.09)
  CFB at Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 8 Hours Postdose | 0.0 (1.52)
  CFB at Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 12 Hours Postdose | 0.0 (1.84)
  CFB at Day 6 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 14 Hours Postdose | -0.4 (1.79)
  CFB at Day 6 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 16 Hours Postdose | 0.1 (2.27)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | 0.3 (1.38)
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | -1.4 (2.28)
  CFB at Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 2 Hours Postdose | -0.4 (2.92)
  CFB at Day 7 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 3 Hours Postdose | -0.5 (2.50)
  CFB at Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 4 Hours Postdose | 0.4 (1.45)
  CFB at Day 7 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 6 Hours Postdose | 0.3 (0.99)
  CFB at Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 8 Hours Postdose | 0.3 (1.33)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | 0.3 (1.94)
  CFB at Day 7 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 14 Hours Postdose | 0.3 (1.59)
  CFB at Day 7 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 16 Hours Postdose | 0.2 (1.76)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.3 (1.27)
  CFB at Day 14 (Follow-up) | 0.5 (1.77)

50. Primary Outcome: CFB in Electrocardiogram (ECG) Mean Heart Rate - Part A
Description: ECG measures included ECG mean heart rate, aggregate PR interval, aggregate RR interval, aggregate QT interval, aggregate QRS duration and aggregate QTcF interval. Baseline is the last measurement taken before the first dose of study drug. L/C indicated levodopa/carbidopa. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
beats/min
  Baseline | 64.7 (11.85)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -0.5 (6.77)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 1.3 (6.78)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | 6.9 (7.65)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 7.1 (8.89)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | 2.5 (5.53)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | 8.2 (5.31)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | 9.0 (10.71)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | 3.7 (4.50)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | 5.9 (7.11)
  Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 6 (SAGE-217): 12 Hours Postdose | 8.5 (5.37)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | 5.9 (8.76)
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | 6.2 (6.03)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | 10.7 (6.78)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.9 (4.17)
  CFB at Day 14 (Follow-up) | 4.7 (9.32)

51. Primary Outcome: CFB in Aggregate PR Interval - Part A
Description: as for outcome 50
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: milliseconds (msec)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
milliseconds (msec)
  Baseline | 158.0 [122 to 228]
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | 2.0 [-16 to 26]
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | -2.0 [-9 to 17]
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | -2.0 [-20 to 25]
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | -8.0 [-26 to 22]
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | -1.0 [-18 to 13]
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -6.0 [-24 to 17]
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | -1.0 [-32 to 18]
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -3.0 [-18 to 21]
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | -5.0 [-25 to 22]
  Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 6 (SAGE-217): 12 Hours Postdose | -1.5 [-30 to 15]
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | -1.0 [-26 to 14]
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | -2.5 [-32 to 19]
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | -2.0 [-18 to 20]
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -2.5 [-24 to 20]
  CFB at Day 14 (Follow-up) | -8.0 [-34 to 86]

52. Primary Outcome: CFB in Aggregate RR Interval - Part A
Description: as for outcome 50
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: milliseconds (msec)
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
milliseconds (msec)
  Baseline | 950.0 [684 to 1226]
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -32.5 [-298 to 190]
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | -43.5 [-298 to 285]
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | -99.0 [-263 to 98]
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | -98.5 [-376 to 252]
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | -56.0 [-143 to 211]
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -102.0 [-276 to -30]
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | -133.0 [-386 to 182]
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -65.0 [-150 to 84]
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | -63.0 [-196 to 36]
  Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 6 (SAGE-217): 12 Hours Postdose | -113.5 [-228 to 28]
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | -76.5 [-420 to 179]
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | -104.5 [-226 to 125]
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | -120.0 [-344 to 70]
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -10.0 [-118 to 114]
  CFB at Day 14 (Follow-up) | -86.0 [-189 to 169]

53. Primary Outcome: CFB in Aggregate QT Interval - Part A
Description: as for outcome 50
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: msec
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
msec
  Baseline | 406.0 [340 to 445]
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -4.0 [-16 to 64]
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | -4.5 [-39 to 39]
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | -9.0 [-44 to 66]
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | -15.5 [-92 to 84]
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | -8.5 [-41 to 22]
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | -12.0 [-42 to 24]
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | -22.0 [-42 to 18]
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -4.5 [-33 to 30]
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | -9.0 [-61 to 9]
  Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 6 (SAGE-217): 12 Hours Postdose | -13.0 [-35 to 26]
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | -12.5 [-48 to 56]
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | -13.0 [-50 to 20]
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | -23.0 [-50 to 55]
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | 0.0 [-26 to 32]
  CFB at Day 14 (Follow-up) | -16.0 [-38 to 20]

54. Primary Outcome: CFB in Aggregate QRS Duration - Part A
Description: as for outcome 50
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: msec
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
msec
  Baseline | 88.0 [76 to 106]
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -1.0 [-14 to 8]
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 0.0 [-5 to 22]
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | 2.0 [-16 to 18]
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 0.0 [-20 to 16]
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | -2.0 [-18 to 16]
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | 0.0 [-14 to 12]
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | -1.0 [-6 to 8]
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | -2.0 [-16 to 15]
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | -0.5 [-18 to 12]
  Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 6 (SAGE-217): 12 Hours Postdose | 0.0 [-14 to 21]
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | -2.0 [-16 to 14]
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | 0.0 [-22 to 14]
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | -1.5 [-12 to 13]
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -1.0 [-16 to 18]
  CFB at Day 14 (Follow-up) | 3.0 [-10 to 12]

55. Primary Outcome: CFB in Aggregate QTcF Interval - Part A
Description: as for outcome 50
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: msec
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
msec
  Baseline | 419.0 [386 to 435]
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | -1.0 [-21 to 39]
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 2.0 [-32 to 33]
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | -0.5 [-29 to 53]
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 6.5 [-85 to 50]
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | -3.0 [-65 to 28]
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | 2.0 [-19 to 31]
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | -7.0 [-23 to 26]
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | 4.5 [-20 to 24]
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | 0.5 [-38 to 32]
  Day 6 (SAGE-217): 12 hours postdose: number analyzed (Participants) | 14
  Day 6 (SAGE-217): 12 hours postdose | -2.5 [-14 to 34]
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | 2.0 [-16 to 32]
  CFB at Day 7 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 Hour Postdose | 0.0 [-35 to 23]
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | -2.5 [-17 to 46]
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -0.5 [-19 to 37]
  CFB at Day 14 (Follow-up) | -7.0 [-52 to 35]

56. Primary Outcome: CFB in Stanford Sleepiness Scale (SSS) Score - Part A
Description: The SSS was a participant-rated scale designed to quickly assess how alert a participant was feeling. Degrees of sleepiness and alertness were rated on a scale of one to seven, where the lowest score of 'one' indicated the participant was 'feeling active, vital, alert, or wide awake' and the highest score of 'seven' indicated the participant was 'no longer fighting sleep, sleep onset soon; having dream-like thoughts'. A negative change from baseline indicated less sleepiness. A positive change from baseline indicated more sleepiness. Baseline is the last measurement taken before the first dose of study drug. L/C indicated levodopa/carbidopa. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
score on a scale
  Baseline | 1.2 (0.56)
  CFB at Day 1 (L/C): 1 Hour Postdose | -0.1 (0.26)
  CFB at Day 1 (L/C): 2 Hours Postdose | -0.1 (0.26)
  CFB at Day 1 (L/C): 3 Hours Postdose | -0.1 (0.52)
  CFB at Day 1 (L/C): 4 Hours Postdose | 0.0 (0.65)
  CFB at Day 1 (L/C): 6 Hours Postdose | 0.0 (0.76)
  CFB at Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 1 (L/C): 8 Hours Postdose | 0.4 (1.39)
  CFB at Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 1 (L/C): 12 Hours Postdose | 0.2 (0.58)
  CFB at Day 1 (L/C): 14 Hours Postdose: number analyzed (Participants) | 12
  CFB at Day 1 (L/C): 14 Hours Postdose | 0.6 (0.90)
  CFB at Day 1 (L/C): 16 Hours Postdose: number analyzed (Participants) | 12
  CFB at Day 1 (L/C): 16 Hours Postdose | 1.0 (0.85)
  CFB at Day 2 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): Predose | 0.4 (0.74)
  CFB at Day 2 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 1 Hour Postdose | 0.3 (0.73)
  CFB at Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 2 Hours Postdose | 0.2 (0.58)
  CFB at Day 2 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 3 Hours Postdose | 0.5 (1.22)
  CFB at Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 4 Hours Postdose | 0.3 (0.91)
  CFB at Day 2 (L/C): 6 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 2 (L/C): 6 Hours Postdose | 0.5 (1.20)
  CFB at Day 2 (L/C): 8 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 2 (L/C): 8 Hours Postdose | 0.4 (0.96)
  CFB at Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 12 Hours Postdose | 0.3 (0.47)
  CFB at Day 2 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 2 (L/C): 14 Hours Postdose | 0.6 (0.94)
  CFB at Day 2 (L/C): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 2 (L/C): 16 Hours Postdose | 0.7 (0.75)
  CFB at Day 3 (L/C): Predose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): Predose | 0.3 (0.91)
  CFB at Day 3 (L/C): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 1 Hour Postdose | 0.0 (0.68)
  CFB at Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 2 Hours Postdose | 0.3 (0.91)
  CFB at Day 3 (L/C): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 3 Hours Postdose | 0.3 (1.07)
  CFB at Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 4 Hours Postdose | 0.4 (1.15)
  CFB at Day 3 (L/C): 6 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 6 Hours Postdose | 0.2 (0.90)
  CFB at Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 3 (L/C): 8 Hours Postdose | 0.3 (0.85)
  CFB at Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 12 Hours Postdose | 0.4 (1.01)
  CFB at Day 3 (L/C): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 3 (L/C): 14 Hours Postdose | 1.0 (1.18)
  CFB at Day 3 (L/C): 16 Hours Postdose: number analyzed (Participants) | 11
  CFB at Day 3 (L/C): 16 Hours Postdose | 0.7 (0.79)
  CFB at Day 4 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): Predose | 0.3 (0.61)
  CFB at Day 4 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 1 Hour Postdose | 3.2 (2.28)
  CFB at Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 2 Hours Postdose | 2.6 (2.03)
  CFB at Day 4 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 3 Hours Postdose | 2.0 (1.57)
  CFB at Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 4 Hours Postdose | 1.2 (1.63)
  CFB at Day 4 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 6 Hours Postdose | 0.4 (1.01)
  CFB at Day 4 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 8 Hours Postdose | 0.2 (0.93)
  CFB at Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 12 Hours Postdose | 0.2 (0.43)
  CFB at Day 4 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 4 (SAGE-217): 14 Hours Postdose | 0.2 (0.43)
  CFB at Day 4 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 4 (SAGE-217): 16 Hours Postdose | 1.0 (0.82)
  CFB at Day 5 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): Predose | 0.3 (0.47)
  CFB at Day 5 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 1 Hour Postdose | 3.8 (1.79)
  CFB at Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 2 Hours Postdose | 1.8 (1.68)
  CFB at Day 5 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 3 Hours Postdose | 1.1 (1.38)
  CFB at Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 4 Hours Postdose | 0.8 (1.42)
  CFB at Day 5 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 6 Hours Postdose | 0.6 (0.96)
  CFB at Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 8 Hours Postdose | 0.1 (0.47)
  CFB at Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 12 Hours Postdose | 0.2 (0.43)
  CFB at Day 5 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 5 (SAGE-217): 14 Hours Postdose | 0.4 (0.94)
  CFB at Day 5 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 5 (SAGE-217): 16 Hours Postdose | 0.8 (1.07)
  CFB at Day 6 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): Predose | 0.1 (0.73)
  CFB at Day 6 (SAGE-217): 1 Hour Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 1 Hour Postdose | 2.6 (1.74)
  CFB at Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 2 Hours Postdose | 1.8 (1.85)
  CFB at Day 6 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 3 Hours Postdose | 1.6 (2.21)
  CFB at Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 4 Hours Postdose | 1.1 (1.94)
  CFB at Day 6 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 6 Hours Postdose | 0.8 (1.30)
  CFB at Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 8 Hours Postdose | 0.3 (0.91)
  CFB at Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 12 Hours Postdose | 0.2 (0.89)
  CFB at Day 6 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 6 (SAGE-217): 14 Hours Postdose | 0.4 (0.74)
  CFB at Day 6 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 13
  CFB at Day 6 (SAGE-217): 16 Hours Postdose | 0.9 (1.19)
  CFB at Day 7 (SAGE-217): Predose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): Predose | 0.2 (0.58)
  CFB at Day 7 (SAGE-217): 1 hour postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 1 hour postdose | 2.0 (1.66)
  CFB at Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 2 Hours Postdose | 1.3 (1.38)
  CFB at Day 7 (SAGE-217): 3 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 3 Hours Postdose | 0.7 (1.14)
  CFB at Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 4 Hours Postdose | 0.7 (1.33)
  CFB at Day 7 (SAGE-217): 6 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 6 Hours Postdose | 0.1 (0.86)
  CFB at Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 8 Hours Postdose | 0.2 (0.97)
  CFB at Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 12 Hours Postdose | 0.1 (0.83)
  CFB at Day 7 (SAGE-217): 14 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 14 Hours Postdose | 0.4 (1.01)
  CFB at Day 7 (SAGE-217): 16 Hours Postdose: number analyzed (Participants) | 14
  CFB at Day 7 (SAGE-217): 16 Hours Postdose | 0.4 (1.01)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 14
  CFB at Day 8 (Follow-up) | -0.1 (0.62)
  CFB at Day 14 (Follow-up) | -0.1 (0.59)

57. Primary Outcome: Percentage of Participants With a Response of 'Yes' to Any Columbia Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation or Suicidal Behavior Item - Part A
Description: The C-SSRS scale consisted of a baseline evaluation (at screening) that assessed the lifetime experience of participants with suicidal ideation (SI) and suicidal behavior (SB) and a postbaseline evaluation that focused on suicidality since the last study visit. The C-SSRS included "yes" or "no"' responses for assessment of suicidal ideation and behavior as well as numeric ratings for the severity of ideation, if present (from 1 to 5, with 5 being the most severe). The C-SSRS SI items involved wish to be dead, non-specific active suicidal thoughts, active SI with any methods, active SI with some intent and active SI with a specific plan. The C-SSRS SB items involved actual attempt, interrupted attempt, aborted attempt, preparatory acts or behavior, suicidal behavior and suicide. The analysis was performed in participants included in Part A of the study.
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug (SAGE-217 or levodopa).
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
percentage of participants
  Suicidal Ideation: Pre-treatment | 0
  Suicidal Ideation: Post-treatment | 0
  Suicidal Behavior: Pre-treatment | 0
  Suicidal Behavior: Post-treatment | 0

58. Primary Outcome: CFB in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II/III Score - Part B
Description: The modified MDS-UPDRS included 4 scales, with various subscales. Each item was rated from 0 (normal) to 4 (severe). The scales were Part I: nonmotor experiences of daily living (13 items); Part II: motor experiences of daily living (13 items); Part III: motor examination (33 scores based on 18 items [several with right, left or other body distribution scores]); and Part IV: motor complications (6 items). The Part II/III tremor score was calculated as the sum of 5 individual tremor item scores from Part II and Part III. The total score range for Part II/III is 0 to 44. Lower scores represent less symptom severity and higher scores represent more symptom severity. Baseline is the last measurement taken before the first dose of study drug. A negative change from baseline indicates an improvement in symptom severity. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Days 1 to 6 (12 and 23 hours postdose), Day 7 (12 hours postdose), Day 14
Population: The efficacy population included all participants in the safety population who received at least one dose of study drug and had at least one postdose MDS-UPDRS evaluation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
score on a scale
  Baseline | 19.1 (3.75)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | -5.4 (4.52)
  CFB at Dose 1 (SAGE-217): 23 Hours Postdose | -5.9 (5.15)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | -6.5 (5.45)
  CFB at Dose 2 (SAGE-217): 23 Hours Postdose | -6.6 (4.60)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -6.0 (4.51)
  CFB at Dose 3 (SAGE-217): 23 Hours Postdose | -5.9 (5.39)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | -8.0 (5.53)
  CFB at Dose 4 (SAGE-217): 23 Hours Postdose | -7.4 (5.02)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -7.4 (7.81)
  CFB at Dose 5 (SAGE-217): 23 Hours Postdose | -8.0 (5.71)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | -5.2 (6.93)
  CFB at Dose 6 (SAGE-217): 23 Hours Postdose | -8.4 (5.02)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -7.7 (4.63)
  CFB at Day 14 (Follow-up) | -3.7 (4.34)

59. Secondary Outcome: MDS-UPDRS Part III Total Score - Part A
Description: Part III of the MDS-UPDRS assessed 18 motor categories, some of which included right and left measurements: speech, facial expression, kinetic tremor of hands, rest tremor amplitude, postural tremor of hands, rigidity of neck and 4 extremities, finger taps, hand movement, pronation/supination, toe tapping, constancy of rest tremor, leg agility, arising from chair, posture, gait, freezing of gait, postural stability, global spontaneity of movement. Part III total score was calculated as the sum of individual item scores from these categories. Each item was rated from 0 (normal) to 4 (severe). The total score range for Part III is 0 to 132. Lower scores indicate less symptom severity. The analysis was performed in participants included in Part A of the study.
Time Frame: Days 1 to 7 (2, 4, 8, and 12 hours postdose), Day 8 and Day 14
Population: The efficacy population included all participants in the safety population who received at least one dose of study drug and had at least one postdose MDS-UPDRS evaluation. Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Antiparkinsonian Agent(s) Followed by SAGE-217
Number analyzed (Participants) | 15
score on a scale
  Day 1 (L/C): 2 Hours Postdose | 25.4 (9.34)
  Day 1 (L/C): 4 Hours Postdose | 30.0 (10.53)
  Day 1 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  Day 1 (L/C): 8 Hours Postdose | 34.3 (10.83)
  Day 1 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 1 (L/C): 12 Hours Postdose | 35.1 (9.71)
  Day 2 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  Day 2 (L/C): 2 Hours Postdose | 27.1 (9.15)
  Day 2 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  Day 2 (L/C): 4 Hours Postdose | 31.1 (9.65)
  Day 2 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  Day 2 (L/C): 8 Hours Postdose | 35.1 (11.37)
  Day 2 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 2 (L/C): 12 Hours Postdose | 36.1 (11.07)
  Day 3 (L/C): 2 Hours Postdose: number analyzed (Participants) | 14
  Day 3 (L/C): 2 Hours Postdose | 26.5 (10.95)
  Day 3 (L/C): 4 Hours Postdose: number analyzed (Participants) | 14
  Day 3 (L/C): 4 Hours Postdose | 29.0 (10.95)
  Day 3 (L/C): 8 Hours Postdose: number analyzed (Participants) | 14
  Day 3 (L/C): 8 Hours Postdose | 35.2 (10.76)
  Day 3 (L/C): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 3 (L/C): 12 Hours Postdose | 36.2 (11.29)
  Day 4 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 11
  Day 4 (SAGE-217): 2 Hours Postdose | 35.7 (14.57)
  Day 4 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  Day 4 (SAGE-217): 4 Hours Postdose | 30.9 (12.84)
  Day 4 (SAGE-217):8 Hours Postdose: number analyzed (Participants) | 14
  Day 4 (SAGE-217):8 Hours Postdose | 33.4 (11.65)
  Day 4 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 4 (SAGE-217): 12 Hours Postdose | 33.3 (13.19)
  Day 5 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 12
  Day 5 (SAGE-217): 2 Hours Postdose | 33.8 (12.76)
  Day 5 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  Day 5 (SAGE-217): 4 Hours Postdose | 32.4 (12.69)
  Day 5 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  Day 5 (SAGE-217): 8 Hours Postdose | 30.9 (12.02)
  Day 5 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 5 (SAGE-217): 12 Hours Postdose | 33.0 (12.15)
  Day 6 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 13
  Day 6 (SAGE-217): 2 Hours Postdose | 31.5 (11.97)
  Day 6 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 13
  Day 6 (SAGE-217): 4 Hours Postdose | 31.8 (9.66)
  Day 6 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  Day 6 (SAGE-217): 8 Hours Postdose | 32.7 (12.81)
  Day 6 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 6 (SAGE-217): 12 Hours Postdose | 34.5 (11.19)
  Day 7 (SAGE-217): 2 Hours Postdose: number analyzed (Participants) | 14
  Day 7 (SAGE-217): 2 Hours Postdose | 36.4 (12.55)
  Day 7 (SAGE-217): 4 Hours Postdose: number analyzed (Participants) | 14
  Day 7 (SAGE-217): 4 Hours Postdose | 35.8 (11.92)
  Day 7 (SAGE-217): 8 Hours Postdose: number analyzed (Participants) | 14
  Day 7 (SAGE-217): 8 Hours Postdose | 36.0 (11.73)
  Day 7 (SAGE-217): 12 Hours Postdose: number analyzed (Participants) | 14
  Day 7 (SAGE-217): 12 Hours Postdose | 35.6 (11.03)
  Day 8 (Follow-up): number analyzed (Participants) | 14
  Day 8 (Follow-up) | 35.4 (10.54)
  Day 14 (Follow-up) | 30.2 (13.00)

60. Secondary Outcome: CFB in the MDS-UPDRS Part III Total Score - Part B
Description: Part III of the MDS-UPDRS assessed 18 motor categories, some of which included right and left measurements: speech, facial expression, kinetic tremor of hands, rest tremor amplitude, postural tremor of hands, rigidity of neck and 4 extremities, finger taps, hand movement, pronation/supination, toe tapping, constancy of rest tremor, leg agility, arising from chair, posture, gait, freezing of gait, postural stability, global spontaneity of movement. Part III total score was calculated as the sum of the individual item scores from these categories. Each item was rated from 0 (normal) to 4 (severe). The total score range for Part III is 0 to 132. Lower scores represent less symptom severity. A negative change from baseline indicates an improvement in symptom severity. Baseline is the last measurement taken before the first dose of study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Days 1 to 6 (12 and 23 hours postdose), Day 7 (12 hours postdose), Day 14
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
score on a scale
  Baseline | 52.4 (12.00)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | -8.4 (8.74)
  CFB at Dose 1 (SAGE-217): 23 Hours Postdose | -10.8 (9.90)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | -11.6 (12.83)
  CFB at Dose 2 (SAGE-217): 23 Hours Postdose | -13.5 (7.87)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -12.4 (10.51)
  CFB at Dose 3 (SAGE-217): 23 Hours Postdose | -10.9 (9.39)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | -14.3 (12.25)
  CFB at Dose 4 (SAGE-217): 23 Hours Postdose | -14.8 (10.30)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -14.5 (15.52)
  CFB at Dose 5 (SAGE-217): 23 Hours Postdose | -18.1 (10.10)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | -14.8 (11.81)
  CFB at Dose 6 (SAGE-217): 23 Hours Postdose | -19.5 (9.30)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -18.6 (9.51)
  CFB at Day 14 (Follow-up) | -14.5 (10.54)

61. Secondary Outcome: CFB in the MDS-UPDRS Part I Total Score - Part B
Description: Part I of the MDS-UPDRS assessed 13 nonmotor experiences of daily living categories. Part I total score was calculated as the sum of the individual item scores from these categories. The total score range for Part I is 0 to 52. Lower scores indicate less symptom severity. A negative change from baseline indicates an improvement in symptom severity. Baseline is the last measurement taken before the first dose of study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Day 7 (12 hours postdose), Day 14
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
score on a scale
  Baseline | 9.9 (6.33)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -4.7 (6.54)
  CFB at Day 14 (Follow-up) | -3.9 (6.05)

62. Secondary Outcome: CFB in the MDS-UPDRS Part II Total Score - Part B
Description: Part II of the MDS-UPDRS assessed 13 categories of motor experiences of daily living: speech, salivation and drooling, chewing and swallowing, eating tasks, dressing, hygiene, handwriting, doing hobbies and other activities, turning in bed, tremor, getting out of bed, car, or deep chair, walking and balance, and freezing. The Part II total score was calculated as the sum of the individual item scores from these categories. The total score range for Part II is 0 to 52. Lower scores indicate less symptom severity. A negative change from baseline indicates an improvement in symptom severity. Baseline is the last measurement taken before the first dose of study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Days 1 to 6 (12 and 23 hours postdose), Day 7 (12 hours postdose), Day 14
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
score on a scale
  Baseline | 15.1 (8.26)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | -1.9 (3.46)
  CFB at Dose 1 (SAGE-217): 23 Hours Postdose | -1.7 (3.73)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | -2.1 (5.17)
  CFB at Dose 2 (SAGE-217): 23 Hours Postdose | -2.2 (4.92)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -2.0 (5.48)
  CFB at Dose 3 (SAGE-217): 23 Hours Postdose | -3.1 (4.20)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | -3.4 (6.33)
  CFB at Dose 4 (SAGE-217): 23 Hours Postdose | -2.4 (5.43)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -4.6 (5.71)
  CFB at Dose 5 (SAGE-217): 23 Hours Postdose | -2.9 (4.90)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | -2.9 (5.05)
  CFB at Dose 6 (SAGE-217): 23 Hours Postdose | -3.9 (5.40)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -3.9 (4.34)
  CFB at Day 14 (Follow-up) | -3.9 (5.02)

63. Secondary Outcome: CFB in the MDS-UPDRS Part I-IV Total Score - Part B
Description: The MDS-UPDRS assesses nonmotor experiences, motor experiences, motor skills, and motor complication categories. The MDS-UPDRS Part I-IV total score was calculated as the sum of the individual item scores from these categories. The total score range for Part I-IV is 0 to 260. Lower scores indicate less symptom severity. A negative change from baseline indicates an improvement in symptom severity. Baseline is the last measurement taken before the first dose of study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Baseline, Day 7 (12 hours postdose), Day 14
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
score on a scale
  Baseline | 84.6 (24.01)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -30.0 (17.71)
  CFB at Day 14 (Follow-up) | -24.1 (20.75)

64. Secondary Outcome: Percentage of Participants With TEAEs - Part B
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. A TEAE was as an AE that occurred after the first administration of study drug. The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Number; unit: percentage of participants
Groups:
- Part B: Follow-up: Participants received antiparkinsonian agent(s) at normally prescribed dosing schedule for Days 8 to 14.
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217 | Part B: Follow-up
Number analyzed (Participants) | 14 | 14
percentage of participants | 57.1 | 0

65. Secondary Outcome: Percentage of Participants With TEAEs, Graded by Severity - Part B
Description: Severity was assessed according to the following scale: mild (awareness of sign or symptom, but easily tolerated); moderate (discomfort sufficient to cause interference with normal activities); severe (incapacitating, with inability to perform normal activities). The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217 | Part B: Follow-up
Number analyzed (Participants) | 14 | 14
percentage of participants
  Mild | 42.9 | 0
  Moderate | 14.3 | 0
  Severe | 0 | 0

66. Secondary Outcome: CFB in Basophils - Part B
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, reticulocytes and reticulocytes to erythrocytes ratio. Baseline is the last measurement taken before the first dose of the study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
10^9 cells/L
  Baseline | 0.06 (0.074)
  CFB at Dose 4 (SAGE-217): Predose | 0.02 (0.089)
  CFB at Dose 6 (SAGE-217): Predose | 0.02 (0.058)
  CFB at Day 8 (Follow-up) | -0.03 (0.061)
  CFB at Day 14 (Follow-up) | 0.00 (0.055)

67. Secondary Outcome: CFB in Basophils to Leukocytes Ratio (%) - Part B
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets, reticulocytes and reticulocytes to erythrocytes ratio. Baseline is the last measurement taken before the first dose of the study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study. The blood cell differential (ratio) data are presented as SI unit, percentage (%).
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
percentage
  Baseline | 1.0 (0.39)
  CFB at Dose 4 (SAGE-217): Predose | 0.2 (0.97)
  CFB at Dose 6 (SAGE-217): Predose | 0.1 (1.00)
  CFB at Day 8 (Follow-up) | -0.1 (0.47)
  CFB at Day 14 (Follow-up) | 0.1 (0.73)

68. Secondary Outcome: CFB in Eosinophils - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
10^9 cells/L
  Baseline | 0.12 (0.058)
  CFB at Dose 4 (SAGE-217): Predose | 0.05 (0.065)
  CFB at Dose 6 (SAGE-217): Predose | 0.03 (0.083)
  CFB at Day 8 (Follow-up) | 0.03 (0.114)
  CFB at Day 14 (Follow-up) | -0.02 (0.058)

69. Secondary Outcome: CFB in Eosinophils to Leukocytes Ratio (%) - Part B
Description: as for outcome 67
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
percentage
  Baseline | 2.0 (1.04)
  CFB at Dose 4 (SAGE-217): Predose | 0.7 (1.20)
  CFB at Dose 6 (SAGE-217): Predose | 0.1 (0.95)
  CFB at Day 8 (Follow-up) | 0.4 (2.06)
  CFB at Day 14 (Follow-up) | -0.4 (0.93)

70. Secondary Outcome: CFB in Erythrocytes - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
10^12 cells/L
  Baseline | 4.65 (0.335)
  CFB at Dose 4 (SAGE-217): Predose | 0.16 (0.798)
  CFB at Dose 6 (SAGE-217): Predose | -0.11 (0.186)
  CFB at Day 8 (Follow-up) | -0.02 (0.208)
  CFB at Day 14 (Follow-up) | -0.06 (0.101)

71. Secondary Outcome: CFB in Hematocrit - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
L/L
  Baseline | 0.436 (0.0357)
  CFB at Dose 4 (SAGE-217): Predose | 0.023 (0.0775)
  CFB at Dose 6 (SAGE-217): Predose | -0.011 (0.0182)
  CFB at Day 8 (Follow-up) | 0.006 (0.0268)
  CFB at Day 14 (Follow-up) | -0.002 (0.0119)

72. Secondary Outcome: CFB in Hemoglobin - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
g/L
  Baseline | 140.1 (14.22)
  CFB at Dose 4 (SAGE-217): Predose | 4.9 (20.90)
  CFB at Dose 6 (SAGE-217): Predose | -1.4 (5.32)
  CFB at Day 8 (Follow-up) | 1.8 (6.03)
  CFB at Day 14 (Follow-up) | -0.7 (4.48)

73. Secondary Outcome: CFB in Leukocytes - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
10^9 cells/L
  Baseline | 6.47 (1.322)
  CFB at Dose 4 (SAGE-217): Predose | 0.85 (2.677)
  CFB at Dose 6 (SAGE-217): Predose | 0.31 (1.370)
  CFB at Day 8 (Follow-up) | -0.21 (0.935)
  CFB at Day 14 (Follow-up) | 0.29 (1.287)

74. Secondary Outcome: CFB in Lymphocytes - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
10^9 cells/L
  Baseline | 1.68 (0.549)
  CFB at Dose 4 (SAGE-217): Predose | 0.44 (0.857)
  CFB at Dose 6 (SAGE-217): Predose | 0.26 (0.386)
  CFB at Day 8 (Follow-up) | 0.18 (0.283)
  CFB at Day 14 (Follow-up) | 0.11 (0.373)

75. Secondary Outcome: CFB in Lymphocytes to Leukocytes Ratio (%) - Part B
Description: as for outcome 67
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
percentage
  Baseline | 26.0 (6.31)
  CFB at Dose 4 (SAGE-217): Predose | 2.5 (6.15)
  CFB at Dose 6 (SAGE-217): Predose | 2.6 (5.34)
  CFB at Day 8 (Follow-up) | 3.4 (5.57)
  CFB at Day 14 (Follow-up) | 0.6 (5.73)

76. Secondary Outcome: CFB in Monocytes - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
10^9 cells/L
  Baseline | 0.40 (0.096)
  CFB at Dose 4 (SAGE-217): Predose | 0.09 (0.194)
  CFB at Dose 6 (SAGE-217): Predose | 0.03 (0.083)
  CFB at Day 8 (Follow-up) | 0.03 (0.133)
  CFB at Day 14 (Follow-up) | 0.01 (0.110)

77. Secondary Outcome: CFB in Monocytes to Leukocytes Ratio (%) - Part B
Description: as for outcome 67
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
percentage
  Baseline | 6.4 (1.55)
  CFB at Dose 4 (SAGE-217): Predose | 0.3 (1.68)
  CFB at Dose 6 (SAGE-217): Predose | 0.1 (1.49)
  CFB at Day 8 (Follow-up) | 0.4 (1.74)
  CFB at Day 14 (Follow-up) | -0.1 (1.07)

78. Secondary Outcome: CFB in Neutrophils - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
10^9 cells/L
  Baseline | 4.23 (0.957)
  CFB at Dose 4 (SAGE-217): Predose | 0.23 (1.842)
  CFB at Dose 6 (SAGE-217): Predose | 0.00 (1.136)
  CFB at Day 8 (Follow-up) | -0.43 (0.902)
  CFB at Day 14 (Follow-up) | 0.16 (1.153)

79. Secondary Outcome: CFB in Neutrophils to Leukocytes Ratio (%) - Part B
Description: as for outcome 67
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
percentage
  Baseline | 65.3 (5.28)
  CFB at Dose 4 (SAGE-217): Predose | -4.2 (7.50)
  CFB at Dose 6 (SAGE-217): Predose | -3.0 (6.64)
  CFB at Day 8 (Follow-up) | -4.4 (6.69)
  CFB at Day 14 (Follow-up) | -0.4 (6.69)

80. Secondary Outcome: CFB in Platelets - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
10^9 cells/L
  Baseline | 189.2 (37.72)
  CFB at Dose 4 (SAGE-217): Predose | 24.1 (67.75)
  CFB at Dose 6 (SAGE-217): Predose | 5.9 (13.64)
  CFB at Day 8 (Follow-up) | 0.8 (20.01)
  CFB at Day 14 (Follow-up) | 5.3 (19.58)

81. Secondary Outcome: CFB in Reticulocytes - Part B
Description: as for outcome 66
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug. Number analyzed = Number of participants with data available at the specific time point.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
10^9 cells/L
  Baseline | 59.3 (19.27)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 13
  CFB at Dose 4 (SAGE-217): Predose | 1.1 (11.35)
  CFB at Dose 6 (SAGE-217): Predose | 5.1 (19.61)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 12
  CFB at Day 8 (Follow-up) | 2.4 (15.55)
  CFB at Day 14 (Follow-up) | 5.1 (20.99)

82. Secondary Outcome: CFB in Reticulocytes to Erythrocytes Ratio (%) - Part B
Description: as for outcome 67
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
percentage
  Baseline | 1.28 (0.417)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 13
  CFB at Dose 4 (SAGE-217): Predose | 0.04 (0.250)
  CFB at Dose 6 (SAGE-217): Predose | 0.13 (0.410)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 12
  CFB at Day 8 (Follow-up) | 0.05 (0.334)
  CFB at Day 14 (Follow-up) | 0.13 (0.486)

83. Secondary Outcome: CFB in Activated Partial Thromboplastin Time - Part B
Description: Coagulation measures included activated partial thromboplastin time, prothrombin international normalized ratio and prothrombin time. Baseline is the last measurement taken before the first dose of the study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Median (Full Range); unit: sec
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
sec
  Baseline | 25.05 [22.0 to 27.5]
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -0.40 [-2.1 to 0.2]
  CFB at Dose 6 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 6 (SAGE-217): Predose | -0.05 [-1.7 to 1.2]
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | -0.30 [-1.6 to 0.5]
  CFB at Day 14 (Follow-up) | -0.20 [-1.4 to 1.7]

84. Secondary Outcome: CFB in Prothrombin International Normalized Ratio - Part B
Description: as for outcome 83
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
ratio
  Baseline | 0.98 (0.043)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -0.03 (0.045)
  CFB at Dose 6 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 6 (SAGE-217): Predose | -0.01 (0.051)
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | 0.00 (0.041)
  CFB at Day 14 (Follow-up) | 0.01 (0.036)

85. Secondary Outcome: CFB in Prothrombin Time - Part B
Description: as for outcome 83
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Median (Full Range); unit: sec
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
sec
  Baseline | 10.60 [9.6 to 11.0]
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -0.20 [-0.8 to 0.6]
  CFB at Dose 6 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 6 (SAGE-217): Predose | -0.05 [-0.5 to 0.5]
  CFB at Day 8 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 8 (Follow-up) | -0.10 [-0.4 to 0.5]
  CFB at Day 14 (Follow-up) | 0.10 [-0.3 to 0.6]

86. Secondary Outcome: CFB in Alanine Aminotransferase - Part B
Description: Clinical chemistry measures included alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bicarbonate, bilirubin, calcium, chloride, creatinine, lipase, magnesium, phosphate, potassium, protein, sodium, urate and urea nitrogen. Baseline is the last measurement taken before the first dose of the study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
U/L
  Baseline | 10.0 (6.66)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 0.3 (3.17)
  CFB at Dose 6 (SAGE-217): Predose | 2.6 (5.42)
  CFB at Day 8 (Follow-up) | 1.9 (3.79)
  CFB at Day 14 (Follow-up) | -0.2 (3.70)

87. Secondary Outcome: CFB in Albumin - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
g/L
  Baseline | 44.2 (2.75)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -0.2 (1.40)
  CFB at Dose 6 (SAGE-217): Predose | -0.6 (1.65)
  CFB at Day 8 (Follow-up) | 0.16 (1.45)
  CFB at Day 14 (Follow-up) | -0.1 (1.86)

88. Secondary Outcome: CFB in Alkaline Phosphatase - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
U/L
  Baseline | 84.0 (22.05)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 1.4 (7.55)
  CFB at Dose 6 (SAGE-217): Predose | 2.1 (3.23)
  CFB at Day 8 (Follow-up) | 2.2 (8.85)
  CFB at Day 14 (Follow-up) | -1.1 (8.69)

89. Secondary Outcome: CFB in Aspartate Aminotransferase - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
U/L
  Baseline | 17.7 (10.59)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -2.8 (10.63)
  CFB at Dose 6 (SAGE-217): Predose | -1.4 (10.93)
  CFB at Day 8 (Follow-up) | -0.4 (11.51)
  CFB at Day 14 (Follow-up) | -2.4 (10.12)

90. Secondary Outcome: CFB in Bicarbonate - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmol/L
  Baseline | 24.6 (1.74)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -1.2 (1.90)
  CFB at Dose 6 (SAGE-217): Predose | -0.9 (2.06)
  CFB at Day 8 (Follow-up) | -1.1 (2.23)
  CFB at Day 14 (Follow-up) | -0.3 (1.77)

91. Secondary Outcome: CFB in Bilirubin - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
umol/L
  Baseline | 8.306 (2.4050)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -2.993 (2.4320)
  CFB at Dose 6 (SAGE-217): Predose | -2.795 (2.0751)
  CFB at Day 8 (Follow-up) | -0.122 (2.4611)
  CFB at Day 14 (Follow-up) | 0.366 (3.0129)

92. Secondary Outcome: CFB in Calcium - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmol/L
  Baseline | 2.340 (0.0796)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 0.006 (0.0859)
  CFB at Dose 6 (SAGE-217): Predose | 0.002 (0.0599)
  CFB at Day 8 (Follow-up) | 0.023 (0.0638)
  CFB at Day 14 (Follow-up) | -0.027 (0.0709)

93. Secondary Outcome: CFB in Chloride - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmol/L
  Baseline | 102.1 (2.03)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 0.1 (1.38)
  CFB at Dose 6 (SAGE-217): Predose | 0.2 (1.53)
  CFB at Day 8 (Follow-up) | -0.5 (2.10)
  CFB at Day 14 (Follow-up) | -0.2 (2.36)

94. Secondary Outcome: CFB in Creatinine - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
umol/L
  Baseline | 80.381 (23.1753)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 11.345 (17.8035)
  CFB at Dose 6 (SAGE-217): Predose | 2.084 (12.3449)
  CFB at Day 8 (Follow-up) | -2.968 (8.0917)
  CFB at Day 14 (Follow-up) | -0.253 (10.0339)

95. Secondary Outcome: CFB in Lipase - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
U/L
  Baseline | 37.2 (16.74)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 15.4 (9.64)
  CFB at Dose 6 (SAGE-217): Predose | 19.4 (16.88)
  CFB at Day 8 (Follow-up) | 4.3 (6.08)
  CFB at Day 14 (Follow-up) | 1.6 (9.30)

96. Secondary Outcome: CFB in Magnesium - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmol/L
  Baseline | 0.873 (0.0489)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -0.014 (0.0536)
  CFB at Dose 6 (SAGE-217): Predose | -0.009 (0.0401)
  CFB at Day 8 (Follow-up) | 0.018 (0.0448)
  CFB at Day 14 (Follow-up) | -0.012 (0.0591)

97. Secondary Outcome: CFB in Phosphate - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmol/L
  Baseline | 1.091 (0.1489)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 0.161 (0.1496)
  CFB at Dose 6 (SAGE-217): Predose | 0.180 (0.1386)
  CFB at Day 8 (Follow-up) | 0.042 (0.1775)
  CFB at Day 14 (Follow-up) | 0.009 (0.1939)

98. Secondary Outcome: CFB in Potassium - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmol/L
  Baseline | 4.57 (0.292)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 0.03 (0.319)
  CFB at Dose 6 (SAGE-217): Predose | -0.11 (0.264)
  CFB at Day 8 (Follow-up) | -0.11 (0.295)
  CFB at Day 14 (Follow-up) | -0.01 (0.268)

99. Secondary Outcome: CFB in Protein - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
g/L
  Baseline | 69.6 (5.40)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -0.8 (1.75)
  CFB at Dose 6 (SAGE-217): Predose | -0.9 (3.00)
  CFB at Day 8 (Follow-up) | 0.9 (2.68)
  CFB at Day 14 (Follow-up) | -0.1 (3.00)

100. Secondary Outcome: CFB in Sodium - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmol/L
  Baseline | 141.8 (1.97)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 0.1 (1.78)
  CFB at Dose 6 (SAGE-217): Predose | 0.1 (1.46)
  CFB at Day 8 (Follow-up) | 0.4 (2.21)
  CFB at Day 14 (Follow-up) | -0.1 (3.00)

101. Secondary Outcome: CFB in Urate - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmol/L
  Baseline | 0.291 (0.0748)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | -0.001 (0.0252)
  CFB at Dose 6 (SAGE-217): Predose | 0.001 (0.0360)
  CFB at Day 8 (Follow-up) | 0.006 (0.0254)
  CFB at Day 14 (Follow-up) | 0.007 (0.0319)

102. Secondary Outcome: CFB in Urea Nitrogen - Part B
Description: as for outcome 86
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmol/L
  Baseline | 5.993 (1.7667)
  CFB at Dose 4 (SAGE-217): Predose: number analyzed (Participants) | 12
  CFB at Dose 4 (SAGE-217): Predose | 2.142 (1.9554)
  CFB at Dose 6 (SAGE-217): Predose | 1.275 (1.7917)
  CFB at Day 8 (Follow-up) | 0.663 (1.9345)
  CFB at Day 14 (Follow-up) | 0.153 (1.2580)

103. Secondary Outcome: CFB in Specific Gravity - Part B
Description: Urinalysis measures included specific gravity and pH. Baseline is the last measurement taken before the first dose of study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
ratio
  Baseline | 1.018 (0.0061)
  CFB at Dose 4 (SAGE-217): Predose | 0.003 (0.0038)
  CFB at Dose 6 (SAGE-217): Predose | 0.001 (0.0053)
  CFB at Day 8 (Follow-up) | -0.004 (0.0077)
  CFB at Day 14 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 14 (Follow-up) | 0.000 (0.0063)

104. Secondary Outcome: CFB in pH - Part B
Description: as for outcome 103
Time Frame: Day 1 to Day 14
Population: as for outcome 81
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
pH
  Baseline | 6.11 (0.924)
  CFB at Dose 4 (SAGE-217): Predose | -0.18 (1.103)
  CFB at Dose 6 (SAGE-217): Predose | -0.32 (1.085)
  CFB at Day 8 (Follow-up) | 0.39 (0.984)
  CFB at Day 14 (Follow-up): number analyzed (Participants) | 13
  CFB at Day 14 (Follow-up) | -0.12 (0.820)

105. Secondary Outcome: CFB in Temperature - Part B
Description: Vital sign measures included temperature, heart rate, respiratory rate, supine systolic blood pressure, standing systolic blood pressure, supine diastolic blood pressure, standing diastolic blood pressure and pulse oximetry. Baseline is the last measurement taken before the first dose of study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
degrees C
  Baseline | 36.56 (0.306)
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | -0.10 (0.199)
  CFB at Dose 1 (SAGE-217): 2 Hours Postdose | 0.01 (0.316)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | -0.19 (0.316)
  CFB at Dose 2 (SAGE-217): Predose | -0.23 (0.370)
  CFB at Dose 2 (SAGE-217): 1 Hour Postdose | -0.15 (0.375)
  CFB at Dose 2 (SAGE-217): 2 Hours Postdose | -0.03 (0.310)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | -0.09 (0.380)
  CFB at Dose 3 (SAGE-217): Predose | -0.06 (0.485)
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -0.11 (0.327)
  CFB at Dose 3 (SAGE-217): 2 Hours Postdose | -0.15 (0.282)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -0.06 (0.386)
  CFB at Dose 4 (SAGE-217): Predose | -0.10 (0.451)
  CFB at Dose 4 (SAGE-217): 1 Hour Postdose | 0.01 (0.408)
  CFB at Dose 4 (SAGE-217): 2 Hours Postdose | -0.09 (0.358)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | -0.12 (0.336)
  CFB at Dose 5 (SAGE-217): Predose | -0.08 (0.418)
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | -0.08 (0.423)
  CFB at Dose 5 (SAGE-217): 2 Hours Postdose | -0.09 (0.562)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -0.09 (0.512)
  CFB at Dose 6 (SAGE-217): Predose | 0.01 (0.240)
  CFB at Dose 6 (SAGE-217): 1 Hour Postdose | 0.05 (0.266)
  CFB at Dose 6 (SAGE-217): 2 Hours Postdose | -0.05 (0.289)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | -0.07 (0.363)
  CFB at Dose 7 (SAGE-217): Predose | -0.07 (0.477)
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | -0.10 (0.348)
  CFB at Dose 7 (SAGE-217): 2 Hours Postdose | -0.08 (0.352)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -0.10 (0.415)
  CFB at Day 14 (Follow-up) | -0.01 (0.291)

106. Secondary Outcome: CFB in Heart Rate - Part B
Description: as for outcome 105
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
beats/min
  Baseline | 72.9 (9.25)
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | 0.1 (7.82)
  CFB at Dose 1 (SAGE-217): 2 Hours Postdose | 0.1 (7.78)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | -3.6 (15.35)
  CFB at Dose 2 (SAGE-217): Predose | -1.6 (7.14)
  CFB at Dose 2 (SAGE-217): 1 Hour Postdose | 0.4 (12.44)
  CFB at Dose 2 (SAGE-217): 2 Hours Postdose | 2.5 (11.94)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | -3.0 (11.08)
  CFB at Dose 3 (SAGE-217): Predose | 0.3 (9.02)
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -0.1 (7.67)
  CFB at Dose 3 (SAGE-217): 2 Hours Postdose | 3.1 (7.95)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -0.1 (10.36)
  CFB at Dose 4 (SAGE-217): Predose | 2.5 (8.16)
  CFB at Dose 4 (SAGE-217): 1 Hour Postdose | 1.4 (9.41)
  CFB at Dose 4 (SAGE-217): 2 Hours Postdose | 1.4 (8.31)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | -1.6 (9.65)
  CFB at Dose 5 (SAGE-217): Predose | 2.5 (8.97)
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | 1.9 (10.61)
  CFB at Dose 5 (SAGE-217): 2 Hours Postdose | -0.4 (9.08)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -4.1 (9.12)
  CFB at Dose 6 (SAGE-217): Predose | 2.1 (8.61)
  CFB at Dose 6 (SAGE-217): 1 Hour Postdose | 1.6 (7.08)
  CFB at Dose 6 (SAGE-217): 2 Hours Postdose | 1.2 (6.13)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | 2.4 (11.29)
  CFB at Dose 7 (SAGE-217): Predose | -1.7 (8.42)
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | -1.7 (8.76)
  CFB at Dose 7 (SAGE-217): 2 Hours Postdose | 0.9 (8.93)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -1.3 (6.83)
  CFB at Day 14 (Follow-up) | -5.0 (8.34)

107. Secondary Outcome: CFB in Respiratory Rate - Part B
Description: as for outcome 105
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
breaths/min
  Baseline | 15.6 (1.91)
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | 0.6 (1.99)
  CFB at Dose 1 (SAGE-217): 2 Hours Postdose | 0.6 (1.98)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | 0.8 (1.31)
  CFB at Dose 2 (SAGE-217): Predose | -0.9 (2.07)
  CFB at Dose 2 (SAGE-217): 1 Hour Postdose | -0.9 (2.09)
  CFB at Dose 2 (SAGE-217): 2 Hours Postdose | 0.4 (1.50)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | 0.8 (1.58)
  CFB at Dose 3 (SAGE-217): Predose | 0.5 (1.79)
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -0.4 (1.74)
  CFB at Dose 3 (SAGE-217): 2 Hours Postdose | -0.6 (2.03)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | 0.6 (1.50)
  CFB at Dose 4 (SAGE-217): Predose | -0.2 (2.36)
  CFB at Dose 4 (SAGE-217): 1 Hour Postdose | -0.4 (1.55)
  CFB at Dose 4 (SAGE-217): 2 Hours Postdose | -0.3 (1.86)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | 1.4 (1.87)
  CFB at Dose 5 (SAGE-217): Predose | 0.4 (1.45)
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | 1.4 (1.98)
  CFB at Dose 5 (SAGE-217): 2 Hours Postdose | 0.6 (2.38)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | 0.4 (1.79)
  CFB at Dose 6 (SAGE-217): Predose | 0.4 (1.74)
  CFB at Dose 6 (SAGE-217): 1 Hour Postdose | -0.1 (1.64)
  CFB at Dose 6 (SAGE-217): 2 Hours Postdose | 0.5 (1.99)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | 0.4 (1.78)
  CFB at Dose 7 (SAGE-217): Predose | -1.1 (2.02)
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | 1.6 (1.39)
  CFB at Dose 7 (SAGE-217): 2 Hours Postdose | -0.7 (2.40)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | 0.6 (1.65)
  CFB at Day 14 (Follow-up) | 0.3 (1.90)

108. Secondary Outcome: CFB in Supine Systolic Blood Pressure - Part B
Description: as for outcome 105
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmHg
  Baseline | 131.7 (16.50)
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | -1.7 (9.15)
  CFB at Dose 1 (SAGE-217): 2 Hours Postdose | -1.4 (7.60)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | 0.3 (13.81)
  CFB at Dose 2 (SAGE-217): Predose | -3.3 (18.20)
  CFB at Dose 2 (SAGE-217): 1 Hour Postdose | 2.9 (14.61)
  CFB at Dose 2 (SAGE-217): 2 Hours Postdose | 0.1 (16.11)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | 6.1 (18.57)
  CFB at Dose 3 (SAGE-217): Predose | -1.2 (12.35)
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -0.1 (10.64)
  CFB at Dose 3 (SAGE-217): 2 Hours Postdose | -1.6 (13.21)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -1.1 (22.03)
  CFB at Dose 4 (SAGE-217): Predose | -1.4 (16.26)
  CFB at Dose 4 (SAGE-217): 1 Hour Postdose | -1.1 (14.22)
  CFB at Dose 4 (SAGE-217): 2 Hours Postdose | -4.3 (14.21)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | 1.2 (18.07)
  CFB at Dose 5 (SAGE-217): Predose | -5.7 (14.67)
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | -4.0 (15.54)
  CFB at Dose 5 (SAGE-217): 2 Hours Postdose | -3.6 (18.79)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | 2.3 (11.82)
  CFB at Dose 6 (SAGE-217): Predose | -10.9 (17.18)
  CFB at Dose 6 (SAGE-217): 1 Hour Postdose | -6.5 (18.68)
  CFB at Dose 6 (SAGE-217): 2 Hours Postdose | -2.8 (18.48)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | -4.1 (15.90)
  CFB at Dose 7 (SAGE-217): Predose | -1.7 (12.63)
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | 2.4 (12.33)
  CFB at Dose 7 (SAGE-217): 2 Hours Postdose | 2.5 (11.94)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -1.2 (13.98)
  CFB at Day 14 (Follow-up) | 3.4 (15.55)

109. Secondary Outcome: CFB in Standing Systolic Blood Pressure - Part B
Description: as for outcome 105
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmHg
  Baseline | 127.8 (14.89)
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | -2.9 (10.51)
  CFB at Dose 1 (SAGE-217): 2 Hours Postdose | -2.4 (8.41)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | 0.6 (7.68)
  CFB at Dose 2 (SAGE-217): Predose | -3.4 (15.96)
  CFB at Dose 2 (SAGE-217): 1 Hour Postdose | -1.5 (14.03)
  CFB at Dose 2 (SAGE-217): 2 Hours Postdose | 1.7 (15.49)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | -0.8 (13.50)
  CFB at Dose 3 (SAGE-217): Predose | -4.2 (11.77)
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -0.8 (11.56)
  CFB at Dose 3 (SAGE-217): 2 Hours Postdose | -4.4 (11.21)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | 0.0 (17.29)
  CFB at Dose 4 (SAGE-217): Predose | -4.5 (12.68)
  CFB at Dose 4 (SAGE-217): 1 Hour Postdose | -4.1 (18.50)
  CFB at Dose 4 (SAGE-217): 2 Hours Postdose | -5.5 (11.25)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | -3.8 (13.38)
  CFB at Dose 5 (SAGE-217): Predose | -7.5 (8.26)
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | -3.9 (12.07)
  CFB at Dose 5 (SAGE-217): 2 Hours Postdose | -5.6 (14.59)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -2.3 (10.01)
  CFB at Dose 6 (SAGE-217): Predose | -9.4 (8.80)
  CFB at Dose 6 (SAGE-217): 1 Hour Postdose | -6.6 (11.05)
  CFB at Dose 6 (SAGE-217): 2 Hours Postdose | -4.7 (10.25)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | -8.6 (11.05)
  CFB at Dose 7 (SAGE-217): Predose | -1.2 (9.01)
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | 1.4 (10.60)
  CFB at Dose 7 (SAGE-217): 2 Hours Postdose | 3.5 (13.18)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -7.5 (12.79)
  CFB at Day 14 (Follow-up) | 0.7 (14.50)

110. Secondary Outcome: CFB in Supine Diastolic Blood Pressure - Part B
Description: as for outcome 105
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmHg
  Baseline | 78.2 (7.49)
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | 0.7 (7.13)
  CFB at Dose 1 (SAGE-217): 2 Hours Postdose | 1.6 (7.20)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | 0.6 (7.23)
  CFB at Dose 2 (SAGE-217): Predose | -0.1 (10.00)
  CFB at Dose 2 (SAGE-217): 1 Hour Postdose | 1.9 (9.23)
  CFB at Dose 2 (SAGE-217): 2 Hours Postdose | -0.5 (9.75)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | 1.9 (9.07)
  CFB at Dose 3 (SAGE-217): Predose | 0.1 (8.54)
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -1.4 (7.39)
  CFB at Dose 3 (SAGE-217): 2 Hours Postdose | -0.9 (12.21)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | 0.6 (11.15)
  CFB at Dose 4 (SAGE-217): Predose | -0.3 (9.24)
  CFB at Dose 4 (SAGE-217): 1 Hour Postdose | 1.5 (8.29)
  CFB at Dose 4 (SAGE-217): 2 Hours Postdose | 0.3 (8.18)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | 0.4 (9.76)
  CFB at Dose 5 (SAGE-217): Predose | -1.1 (9.05)
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | -0.7 (9.92)
  CFB at Dose 5 (SAGE-217): 2 Hours Postdose | -0.6 (9.44)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -0.6 (9.00)
  CFB at Dose 6 (SAGE-217): Predose | -2.4 (9.24)
  CFB at Dose 6 (SAGE-217): 1 Hour Postdose | 1.1 (9.49)
  CFB at Dose 6 (SAGE-217): 2 Hours Postdose | 0.6 (9.15)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | 1.9 (9.74)
  CFB at Dose 7 (SAGE-217): Predose | -0.6 (9.16)
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | 1.8 (10.50)
  CFB at Dose 7 (SAGE-217): 2 Hours Postdose | 0.2 (8.50)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | 0.4 (8.93)
  CFB at Day 14 (Follow-up) | 0.3 (8.30)

111. Secondary Outcome: CFB in Standing Diastolic Blood Pressure - Part B
Description: as for outcome 105
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
mmHg
  Baseline | 81.9 (6.99)
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | -2.0 (6.04)
  CFB at Dose 1 (SAGE-217): 2 Hours Postdose | -2.4 (6.32)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | -1.6 (7.17)
  CFB at Dose 2 (SAGE-217): Predose | -3.9 (7.18)
  CFB at Dose 2 (SAGE-217): 1 Hour Postdose | -2.4 (5.11)
  CFB at Dose 2 (SAGE-217): 2 Hours Postdose | -1.5 (7.69)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | -1.9 (8.64)
  CFB at Dose 3 (SAGE-217): Predose | -3.9 (8.60)
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -1.4 (9.08)
  CFB at Dose 3 (SAGE-217): 2 Hours Postdose | -1.1 (7.44)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -2.4 (7.79)
  CFB at Dose 4 (SAGE-217): Predose | -2.4 (7.53)
  CFB at Dose 4 (SAGE-217): 1 Hour Postdose | -4.1 (9.77)
  CFB at Dose 4 (SAGE-217): 2 Hours Postdose | -2.9 (8.69)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | -2.8 (9.18)
  CFB at Dose 5 (SAGE-217): Predose | -5.5 (8.93)
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | -1.4 (7.91)
  CFB at Dose 5 (SAGE-217): 2 Hours Postdose | -3.1 (8.51)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | 0.0 (10.03)
  CFB at Dose 6 (SAGE-217): Predose | -4.0 (7.74)
  CFB at Dose 6 (SAGE-217): 1 Hour Postdose | -1.6 (8.35)
  CFB at Dose 6 (SAGE-217): 2 Hours Postdose | -2.0 (7.65)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | -2.1 (8.27)
  CFB at Dose 7 (SAGE-217): Predose | -1.7 (9.21)
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | -0.2 (8.86)
  CFB at Dose 7 (SAGE-217): 2 Hours Postdose | 0.6 (8.14)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -2.7 (8.59)
  CFB at Day 14 (Follow-up) | -1.1 (9.21)

112. Secondary Outcome: CFB in Pulse Oximetry - Part B
Description: as for outcome 105
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
percentage
  Baseline | 96.9 (1.51)
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | -0.6 (1.60)
  CFB at Dose 1 (SAGE-217): 2 Hours Postdose | 0.0 (2.08)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | 0.4 (1.86)
  CFB at Dose 2 (SAGE-217): Predose | -0.3 (1.77)
  CFB at Dose 2 (SAGE-217): 1 Hour Postdose | 0.1 (1.64)
  CFB at Dose 2 (SAGE-217): 2 Hours Postdose | 0.1 (1.73)
  CFB at Dose 2 (SAGE-217): 12 Hours Postdose | 0.3 (1.38)
  CFB at Dose 3 (SAGE-217): Predose | 0.1 (1.51)
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | 0.3 (2.02)
  CFB at Dose 3 (SAGE-217): 2 Hours Postdose | -0.5 (1.87)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | 0.0 (2.15)
  CFB at Dose 4 (SAGE-217): Predose | -0.6 (1.69)
  CFB at Dose 4 (SAGE-217): 1 Hour Postdose | 0.6 (1.01)
  CFB at Dose 4 (SAGE-217): 2 Hours Postdose | 0.1 (1.46)
  CFB at Dose 4 (SAGE-217): 12 Hours Postdose | -0.3 (2.09)
  CFB at Dose 5 (SAGE-217): Predose | 0.5 (1.34)
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | 0.6 (1.91)
  CFB at Dose 5 (SAGE-217): 2 Hours Postdose | 0.0 (1.66)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | 0.4 (1.55)
  CFB at Dose 6 (SAGE-217): Predose | -0.2 (1.63)
  CFB at Dose 6 (SAGE-217): 1 Hour Postdose | 0.1 (1.33)
  CFB at Dose 6 (SAGE-217): 2 Hours Postdose | 0.1 (1.33)
  CFB at Dose 6 (SAGE-217): 12 Hours Postdose | 0.3 (1.64)
  CFB at Dose 7 (SAGE-217): Predose | 0.2 (1.25)
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | -0.4 (1.65)
  CFB at Dose 7 (SAGE-217): 2 Hours Postdose | 0.0 (1.71)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | 0.1 (1.79)
  CFB at Day 14 (Follow-up) | 0.5 (1.91)

113. Secondary Outcome: CFB in ECG Mean Heart Rate - Part B
Description: ECG measures included ECG mean heart rate, aggregate PR interval, aggregate RR interval, aggregate QT interval, aggregate QRS duration and aggregate QTcF interval. Baseline is the last measurement taken before the first dose of study drug. Doses 1 to 7 were given on Days 1 to 7, respectively. The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
beats/min
  Baseline | 71.4 (10.24)
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | 0.1 (5.55)
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | -6.6 (7.81)
  CFB at Dose 3 (SAGE-217): Predose | 0.2 (6.19)
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -0.3 (5.03)
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -1.6 (9.88)
  CFB at Dose 5 (SAGE-217): Predose | 2.2 (6.28)
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | 1.8 (7.82)
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -2.4 (9.39)
  CFB at Dose 7 (SAGE-217): Predose | 0.2 (6.81)
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | -0.7 (6.97)
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | 1.4 (6.35)
  CFB at Day 14 (Follow-up) | -6.1 (8.57)

114. Secondary Outcome: CFB in Aggregate PR Interval - Part B
Description: as for outcome 113
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
msec
  Baseline | 174.0 [141 to 203]
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | 2.5 [-20 to 96]
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | 0.0 [-24 to 17]
  CFB at Dose 3 (SAGE-217): Predose | -2.0 [-29 to 8]
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -1.5 [-33 to 8]
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | 3.5 [-27 to 20]
  CFB at Dose 5 (SAGE-217): Predose | 1.5 [-28 to 46]
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | 2.0 [-19 to 12]
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -1.5 [-22 to 22]
  CFB at Dose 7 (SAGE-217): Predose | -2.0 [-17 to 18]
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | 0.0 [-36 to 10]
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -1.5 [-26 to 27]
  CFB at Day 14 (Follow-up) | -2.5 [-31 to 7]

115. Secondary Outcome: CFB in Aggregate RR Interval - Part B
Description: as for outcome 113
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
msec
  Baseline | 823.0 [683 to 1239]
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | -19.0 [-93 to 142]
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | 67.5 [-68 to 366]
  CFB at Dose 3 (SAGE-217): Predose | -32.5 [-85 to 141]
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | -10.0 [-140 to 143]
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | 7.0 [-164 to 231]
  CFB at Dose 5 (SAGE-217): Predose | -23.5 [-132 to 99]
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | -24.5 [-148 to 96]
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | 50.0 [-185 to 304]
  CFB at Dose 7 (SAGE-217): Predose | -16.0 [-80 to 212]
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | -26.0 [-76 to 180]
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | 16.5 [-148 to 74]
  CFB at Day 14 (Follow-up) | 66.0 [-76 to 397]

116. Secondary Outcome: CFB in Aggregate QT Interval - Part B
Description: as for outcome 113
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
msec
  Baseline | 374.0 [361 to 442]
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | 3.5 [-41 to 36]
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | 10.0 [-20 to 70]
  CFB at Dose 3 (SAGE-217): Predose | 2.0 [-21 to 32]
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | 3.5 [-34 to 31]
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | 0.0 [-52 to 31]
  CFB at Dose 5 (SAGE-217): Predose | -1.0 [-35 to 17]
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | -5.5 [-37 to 25]
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | 11.0 [-45 to 41]
  CFB at Dose 7 (SAGE-217): Predose | -5.0 [-23 to 21]
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | 3.5 [-32 to 32]
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | 2.5 [-30 to 21]
  CFB at Day 14 (Follow-up) | 14.0 [-19 to 57]

117. Secondary Outcome: CFB in Aggregate QRS Duration - Part B
Description: as for outcome 113
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
msec
  Baseline | 99.5 [76 to 153]
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | 0.0 [-9 to 12]
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | -1.0 [-8 to 16]
  CFB at Dose 3 (SAGE-217): Predose | -1.5 [-11 to 9]
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | 0.0 [-12 to 10]
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -0.5 [-14 to 6]
  CFB at Dose 5 (SAGE-217): Predose | -1.5 [-10 to 16]
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | 1.5 [-5 to 11]
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | -3.5 [-12 to 6]
  CFB at Dose 7 (SAGE-217): Predose | -0.5 [-5 to 238]
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | -1.0 [-10 to 6]
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | -1.0 [-11 to 6]
  CFB at Day 14 (Follow-up) | 0.5 [-11 to 11]

118. Secondary Outcome: CFB in Aggregate QTcF Interval - Part B
Description: as for outcome 113
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Median (Full Range); unit: msec
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
msec
  Baseline | 407.0 [384 to 432]
  CFB at Dose 1 (SAGE-217): 1 Hour Postdose | 3.0 [-35 to 54]
  CFB at Dose 1 (SAGE-217): 12 Hours Postdose | -2.5 [-34 to 60]
  CFB at Dose 3 (SAGE-217): Predose | 0.0 [-11 to 28]
  CFB at Dose 3 (SAGE-217): 1 Hour Postdose | 0.5 [-18 to 29]
  CFB at Dose 3 (SAGE-217): 12 Hours Postdose | -1.5 [-37 to 12]
  CFB at Dose 5 (SAGE-217): Predose | 1.0 [-19 to 19]
  CFB at Dose 5 (SAGE-217): 1 Hour Postdose | 0.0 [-19 to 22]
  CFB at Dose 5 (SAGE-217): 12 Hours Postdose | 5.5 [-27 to 17]
  CFB at Dose 7 (SAGE-217): Predose | -1.0 [-16 to 29]
  CFB at Dose 7 (SAGE-217): 1 Hour Postdose | -2.0 [-25 to 20]
  CFB at Dose 7 (SAGE-217): 12 Hours Postdose | 2.0 [-11 to 17]
  CFB at Day 14 (Follow-up) | 0.5 [-10 to 21]

119. Secondary Outcome: Percentage of Participants With a Response of 'Yes' to Any C-SSRS Suicidal Ideation or Suicidal Behavior Item - Part B
Description: The C-SSRS scale consisted of a baseline evaluation (at screening) that assessed the lifetime experience of participants with suicidal ideation (SI) and suicidal behavior (SB) and a postbaseline evaluation that focused on suicidality since the last study visit. The C-SSRS included "yes" or "no"' responses for assessment of suicidal ideation and behavior as well as numeric ratings for the severity of ideation, if present (from 1 to 5, with 5 being the most severe). The C-SSRS SI items involved wish to be dead, non-specific active suicidal thoughts, active SI with any methods, active SI with some intent and active SI with a specific plan. The C-SSRS SB items involved actual attempt, interrupted attempt, aborted attempt, preparatory acts or behavior, suicidal behavior and suicide. The analysis was performed in participants included in Part B of the study.
Time Frame: Day 1 to Day 14
Population: The safety population included all participants who were administered study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Antiparkinsonian Agent(s) + SAGE-217
Number analyzed (Participants) | 14
percentage of participants
  Suicidal Ideation: Wish to be Dead: Pre-treatment | 14.3
  Suicidal Ideation: Wish to be Dead: Post-treatment | 0
  Suicidal Behavior: Pre-treatment | 0
  Suicidal Behavior: Post-treatment | 0

ADVERSE EVENTS:
Time Frame: Part A: Up to 14 days; Part B: Up to 14 days
Description: The safety population included all participants who were administered study drug [SAGE-217 or levodopa (Part A); or SAGE-217 or antiparkinsonian agent(s) (Part B)]. Number of participants at risk is number of participants in the safety population that remained in the study during each period.
Groups:
- Part B: SAGE-217 Dose 1 to Dose 7: Participants on a stable dose of antiparkinsonian agent(s) received SAGE-217, up to 30 mg per day, capsules, for Days 1 to 7 in the evening with food.
Arm/Group | Part A: Antiparkinsonian Agent(s) Day 1 to Day 3 | Part A: SAGE-217 Day 4 to Day 7 | Part A: Follow-up | Part B: SAGE-217 Dose 1 to Dose 7 | Part B: Follow-up
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/15 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/15 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 4/15 | 14/14 | 2/15 | 8/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Antiparkinsonian Agent(s) Day 1 to Day 3 (N=15) | Part A: SAGE-217 Day 4 to Day 7 (N=14) | Part A: Follow-up (N=15) | Part B: SAGE-217 Dose 1 to Dose 7 (N=14) | Part B: Follow-up (N=14)
Sedation (Nervous system disorders) | 1 | 10 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 6 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 0 | 2 | 0
Myoclonus (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine with Aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Parkinson's Disease (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Feeling drunk (General disorders) | 0 | 4 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Lipase Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Panic Attack (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (3):
  • Study Protocol (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03000569/Prot_001.pdf
  • Statistical Analysis Plan: Version 2 (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT03000569/SAP_000.pdf
  • Statistical Analysis Plan: Version 1 (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT03000569/SAP_002.pdf